CLINICAL TRIAL: NCT03071692
Title: Pemafibrate to Reduce Cardiovascular OutcoMes by Reducing Triglycerides IN patiENts With diabeTes (PROMINENT)
Acronym: PROMINENT
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was stopped for futility based on efficacy results at the interim analysis; no unexpected safety findings were observed.
Sponsor: Kowa Research Institute, Inc. (Industry)
Collaborators: Brigham and Women's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: K-877-302
Record Dates: First submitted 2017-02-23; First posted 2017-03-07 (Actual); Results first posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Type2 Diabetes; Dyslipidemia
MeSH Terms: conditions — Dyslipidemias | interventions — K-877 compound; (R)-2-(3-((benzoxazol-2-yl-d4 (3-(4-methoxyphenoxy-d7)propyl)amino)methyl)phenoxy) butanoic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): K-877 (pemafibrate) tablet twice daily.
  Interventions: Drug: K-877
- Control Group (Placebo Comparator): Matching K-877 placebo tablet twice daily.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: K-877 — 0.2mg tablet
  Other Names: pemafibrate
  Arms: Treatment Group
Drug: Placebo — K-877 matching placebo tablet
  Arms: Control Group

SUMMARY:
The primary objective of the study is to determine whether pemafibrate administered twice daily will delay the time to first occurrence of any component of the clinical composite endpoint of:

* nonfatal Myocardial Infarction (MI)
* nonfatal ischemic stroke
* coronary revascularization; or
* Cardio Vascular (CV) death.

DETAILED DESCRIPTION:
A multi-regional clinical trial with participating sites in the following countries. India is being conducted under a previous protocol version due to regulatory requirements.

* Argentina
* Brazil
* Bulgaria
* Canada
* Colombia
* Czech Republic
* Denmark
* France
* Germany
* Hungary
* India
* Israel
* Japan
* Mexico
* Netherlands
* Poland
* Romania
* Russian Federation
* Slovakia
* South Africa
* Spain
* Ukraine
* United Kingdom
* United States

ELIGIBILITY:
Inclusion Criteria:

1. Fasting TG ≥ 200 mg/dL (2.26 mmol/L) and < 500 mg/dL (5.65 mmol/L) at Visit 1 (Screening/Enrollment Visit) or Visit 1.1 (Retest)
2. HDL-C ≤ 40 mg/dL (1.03 mmol/L) at Visit 1 (Screening/Enrollment Visit) or Visit 1.1 (Retest)
3. Type 2 diabetes of longer than 12 weeks duration documented in medical records, for example: local laboratory evidence through medical record review of elevated HbA1c (≥ 6.5% [48 mmol/mol]), elevated plasma glucose (fasting ≥ 126 mg/dL [7.0 mmol/L], 2-hour ≥ 200 mg/dL [11.1 mmol/L] during oral glucose tolerance testing, or random value ≥ 200 mg/dL with classic symptoms, or currently taking medication for treatment of diabetes; AND either

   1. Age ≥ 50 years if male or ≥ 55 years if female (primary prevention cohort); OR
   2. Age ≥ 18 years and established systemic atherosclerosis (secondary prevention cohort), defined as any 1 of the following:

      * i. Prior MI or ischemic (non-hemorrhagic) stroke
      * ii. Coronary angiographic lesion of ≥ 60% stenosis in a major epicardial vessel or ≥ 50% left main stenosis
      * iii. Asymptomatic carotid disease with ≥ 70% carotid artery stenosis
      * iv. Symptomatic carotid disease with ≥ 50% carotid artery stenosis
      * v. Symptomatic lower extremity PAD (ie, intermittent claudication, rest pain, lower extremity ischemic ulceration, or major amputation with either ankle-brachial index ≤ 0.9 or other diagnostic testing [eg, toe-brachial index, angiogram, or other imaging study])
      * vi. Prior arterial revascularization procedure (including coronary, carotid, or peripheral angioplasty/stenting, bypass, or atherectomy/endarterectomy)

Exclusion Criteria:

1. Current or planned use of fibrates or agents with PPAR-α agonist activity (eg, saroglitazar) within 6 weeks (42 days) of Visit 1 (Screening/Enrollment Visit). Note: PPAR-γ agonists (eg, glizatones such as pioglitazone and rosiglitazone) are allowed
2. Known sensitivity to PPAR-α agonists or tablet excipients
3. Initiation of, or change in, current TG-lowering therapy within 12 weeks of Visit 1 (if applicable). Note: TG-lowering therapy is defined as niacin > 100 mg/day or dietary supplements or prescription omega-3 fatty acids > 1 g/day
4. Type 1 diabetes mellitus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10544 (Actual)
Dates: Start 2017-03-23 (Actual); Primary Completion 2022-07-27 (Actual); Study Completion 2022-07-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Ridker, MD, Study Director — CCVDP & The Brigham and Women's Hospital; Aruna Pradhan, MD, Study Director — CCVDP & The Brigham and Women's Hospital
Locations (887):
- United States (242):
  - Synexus Clinical Research US, Inc., Birmingham, Alabama
  - University of Alabama at Birmingham, Birmingham, Alabama
  - VA Medical Center - Birmingham, Birmingham, Alabama
  - Alabama Clinical Therapeutics, LLC, Birmingham, Alabama
  - Fundamental Research, LLC, Gulf Shores, Alabama
  - Mobile Heart Specialists, PC, Mobile, Alabama
  - Terence T. Hart, MD, Tuscumbia, Alabama
  - Synexus Clinical Research US, Inc., Chandler, Arizona
  - Synexus Clinical Research US, Inc., Mesa, Arizona
  - Arizona Arthritis & Rheumatology Research, PLLC, Peoria, Arizona
  - Phoenix Veterans Adminstration Health Care System, Phoenix, Arizona
  - Synexus Clinical Research US, Inc., Phoenix, Arizona
  - Clinical Research Institute of Arizona, LLC, Surprise, Arizona
  - Synexus Clinical Research US, Inc., Tucson, Arizona
  - Eclipse Clinical Research, Tucson, Arizona
  - Central Arkansas Veterans Healthcare System, Little Rock, Arkansas
  - Clinical Research Alliance, Inc, Alhambra, California
  - Aurora Care Clinic, Costa Mesa, California
  - AMCR Institute, Inc., Escondido, California
  - National Institute of Clinical Research, Huntington Beach, California
  - VA Loma Linda Healthcare System, Loma Linda, California
  - VA Long Beach Healthcare System, Long Beach, California
  - Eastside Clinical Research Associates, Los Angeles, California
  - VA Greater Los Angeles Healthcare System, Los Angeles, California
  - Richard S. Cherlin, MD, Los Gatos, California
  - Northridge Clinical Research Inc., Northridge, California
  - Palo Alto Division, Palo Alto, California
  - Huntington Hospital - Research Department, Pasadena, California
  - Rancho Cucamonga Clinical Research, Rancho Cucamonga, California
  - MD Strategies Research Centers, San Diego, California
  - Alex Harrison, MD Inc., Santa Maria, California
  - Santa Rosa Cardiology Medical Group, Inc., Santa Rosa, California
  - Blue Coast Cardiology, Vista, California
  - Lynn Institute of Denver, Aurora, Colorado
  - New West Physicians, PC, Golden, Colorado
  - Southwest Family Medicine, Littleton, Colorado
  - Chase Medical Research, LLC, Waterbury, Connecticut
  - VA Connecticut Healthcare Sys, West Haven, Connecticut
  - Cardiology Physicians, PA, Newark, Delaware
  - Bay Pines VA Healthcare System, Bay Pines, Florida
  - Meridien Research, Bradenton, Florida
  - Clinical Research Of Brandon, LLC, Brandon, Florida
  - Clearwater Cardiovascular Consultants, Clearwater, Florida
  - Daytona Heart Group, Daytona Beach, Florida
  - Cohen Medical Research Associates, LLC, Delray Beach, Florida
  - Malcom Randall VA Medical Center, Gainesville, Florida
  - Pines Clinical Research, Inc., Hollywood, Florida
  - Homestead Cardiac & Vein Center, Homestead, Florida
  - Westside Center for Clinical Research, Jacksonville, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Health Awareness, Inc., Jupiter, Florida
  - Meridien Research, Lakeland, Florida
  - Clearwater Cardiovascular & Interventional Consultants, Largo, Florida
  - University of Miami, Miami, Florida
  - Advanced Medical Research Institute, Miami, Florida
  - Ocala Research Institute, Inc., Ocala, Florida
  - Morgan Medical Management & Consultants Inc., Ocala, Florida
  - Endocrine Associates of Florida, Ocoee, Florida
  - Research Physicians Network Alliance, Orlando, Florida
  - Andres Patron, D.O., P.A, Pembroke Pines, Florida
  - DBC Research, Corp, Pembroke Pines, Florida
  - Langhorne Cardiology Consultants, Inc., Pensacola, Florida
  - Clearwater Cardiovascular Consultants, Safety Harbor, Florida
  - Professional Health Care of Pinellas, St. Petersburg, Florida
  - James A. Haley VA Medical Center, Tampa, Florida
  - Clinical Research of Central Florida, Winter Haven, Florida
  - Emory University, Atlanta, Georgia
  - Atlanta Heart Specialists, LLC, Cumming, Georgia
  - VA Medical Center - Atlanta, Decatur, Georgia
  - Alta Pharmaceutical Research Center, Inc., Dunwoody, Georgia
  - Atlanta Heart Specialists, LLC, Tucker, Georgia
  - Christie Clinic, LLC, Champaign, Illinois
  - Apex Medical Research, AMR, Inc., Chicago, Illinois
  - Clinical Investigation Specialists, Inc., Gurnee, Illinois
  - Edward Hines Jr. VA Hospital, Hines, Illinois
  - Advocate Health and Hospitals Corp, Normal, Illinois
  - Captain James A. Lovell Federal Health Care Center, North Chicago, Illinois
  - Specialty Physicians of Illinois, Olympia Fields, Illinois
  - Community Hospital of Anderson and Madison County, Inc., Anderson, Indiana
  - Synexus Clinical Research US, Inc., Evansville, Indiana
  - Deaconess Clinic, Evansville, Indiana
  - VA Medical Center - Indianapolis, Indianapolis, Indiana
  - Cardiovascular Research of Northwest Indiana, LLC, Munster, Indiana
  - Buynak Clinical Research, Valparaiso, Indiana
  - West Broadway Clinic, Council Bluffs, Iowa
  - Iowa Diabetes and Endocrinology Research Center, PLC, Des Moines, Iowa
  - The Iowa Clinic, PC, West Des Moines, Iowa
  - University of Kansas Medical Center Research Institute, Inc., Kansas City, Kansas
  - VA Eastern Kansas Health Care, Leavenworth, Kansas
  - The Research Group of Lexington, LLC, Lexington, Kentucky
  - Robley Rex VA Medical Center, Louisville, Kentucky
  - Cambridge Medical Trials, Alexandria, Louisiana
  - Cardiovascular Associates Research, LLC, Covington, Louisiana
  - Centex Studies Inc., Lake Charles, Louisiana
  - Overton Brooks VA Medical Center, Shreveport, Louisiana
  - Southern Maine Health Care, Biddeford, Maine
  - Baltimore VA medical centre, Baltimore, Maryland
  - University of Maryland School of Medicine, Baltimore, Maryland
  - Maryland Cardiovascular Specialists, Baltimore, Maryland
  - Medstar Health Research Institute, Hyattsville, Maryland
  - Delmarva Heart Research Foundation, Inc., Salisbury, Maryland
  - Joslin Diabetes Center, Boston, Massachusetts
  - Pentucket Medical Associates, Haverhill, Massachusetts
  - South Shore Internal Medicine Associates, Milton, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Veterans Affairs Ann Arbor Healthcare System, Ann Arbor, Michigan
  - Northern Pines Health Center, Buckley, Michigan
  - Cadillac Clinical Research, LLC, Cadillac, Michigan
  - AA MRC LLC Ahmed Arif Medical Research Center, Flint, Michigan
  - Sparrow Clinical Research Institute, Lansing, Michigan
  - Covenant Medical Center, Inc., Saginaw, Michigan
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - Synexus Clinical Research US, Inc., Richfield, Minnesota
  - CentraCare Heart & Vascular, Saint Cloud, Minnesota
  - HealthEast Medical Research Institute, Saint Paul, Minnesota
  - GV Montgomery VA Medical Center, Jackson, Mississippi
  - Kansas City VA Medical Center, Kansas City, Missouri
  - Synexus Clinical Research US, Inc., St Louis, Missouri
  - Kalispell Regional Medical Center dba Glacier View Research Institute, Kalispell, Montana
  - VA Nebraska-Western Iowa Health Care System, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Synexus Clinical Research US, Inc., Papillion, Nebraska
  - Synexus Clinical Research US, Inc., Henderson, Nevada
  - Red Rock Clinical Research LLC, Las Vegas, Nevada
  - VA Sierra Nevada Health Care System, Reno, Nevada
  - Southern New Hampshire Diabetes and Endocrinology, Nashua, New Hampshire
  - Monmouth Cardiology Associates, Eatontown, New Jersey
  - NJ Heart, Linden, New Jersey
  - The Valley Hospital, Ridgewood, New Jersey
  - Raymond G. Murphy VA Medical Center, Albuquerque, New Mexico
  - Endocrine Group, L.L.P., Albany, New York
  - Stratton Veterans Affairs Medical Center - Albany, Albany, New York
  - Buffalo VA Medical Center, Buffalo, New York
  - Winthrop Cardiology Associates, Mineola, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - VA Medical Center - Syracuse, Syracuse, New York
  - Randolph Medical Associates, Asheboro, North Carolina
  - OnSite Clinical Solutions, LLC, Asheville, North Carolina
  - Kernodle Clinic, Inc., Dept. of the Private Diagnostic Clinic, PLLC, Burlington, North Carolina
  - Cary Research Group, LLC, Cary, North Carolina
  - PMG Research of Cary, LLC, Cary, North Carolina
  - Novant Health - Heart and Vascular Institute, Charlotte, North Carolina
  - The Presbyterian Hospital, Charlotte, North Carolina
  - Focus Clinical Research Solutions, Charlotte, North Carolina
  - Medication Management, LLC, Greensboro, North Carolina
  - Triad Clinical Trials, LLC, Greensboro, North Carolina
  - Clinical Trials of America-NC, LLC, Hickory, North Carolina
  - PMG Research of Hickory, LLC, Hickory, North Carolina
  - Research Institute of the Carolinas, PLC, Mooresville, North Carolina
  - Diabetes and Endocrinology Consultants, Morehead City, North Carolina
  - Pinehurst Medical Clinic Inc, Pinehurst, North Carolina
  - PMG Research of Raleigh, LLC, Raleigh, North Carolina
  - PMG Research of Rocky Mount, LLC, Rocky Mount, North Carolina
  - PMG Research of Salisbury, LLC, Salisbury, North Carolina
  - Carolina Research Center, Inc., Shelby, North Carolina
  - Synexus Clinical Research US, Inc., Akron, Ohio
  - OhioHealth Heart & Vascular Physicians (Heartcare, Inc.) - Athens, Athens, Ohio
  - Aultman Hospital, Canton, Ohio
  - Hometown Urgent Care & Occupational Health, Cincinnati, Ohio
  - Cincinnati Veterans Affairs Medical Center, Cincinnati, Ohio
  - Louis Stokes Cleveland Dept of VA Medical Center, Cleveland, Ohio
  - Prestige Clinical Research Center, Franklin, Ohio
  - Craig S Thompson MD LLC, Marion, Ohio
  - Intend Research, Norman, Oklahoma
  - Lynn Institute of Norman, Norman, Oklahoma
  - Oklahoma City Clinic - Central, Oklahoma City, Oklahoma
  - South Oklahoma Heart Research Group, Oklahoma City, Oklahoma
  - Heart Clinic of Southern Oregon, Medford, Oregon
  - Chambersburg Hospital, Chambersburg, Pennsylvania
  - AMH Feasterville Family Health Care Center, Feasterville, Pennsylvania
  - Family Medical Associates, Levittown, Pennsylvania
  - VA Pittsburgh Healthcare System, Pittsburgh, Pennsylvania
  - Preferred Primary Care Physicians, Pittsburgh, Pennsylvania
  - Fay West Family Practice, Scottdale, Pennsylvania
  - Montgomery Medical Inc., Smithfield, Pennsylvania
  - Partners in Clinical Research, Cumberland, Rhode Island
  - Ocean State Clinical Research Partners, Lincoln, Rhode Island
  - Providence Veteran Administration Medical Center, Providence, Rhode Island
  - Synexus Clinical Research US, Inc., Anderson, South Carolina
  - Ralph H. Johnson VA Medical Center, Charleston, South Carolina
  - Mountain View Clinical Research, Inc., Greer, South Carolina
  - Main Street Physician's Care - Waterway, Little River, South Carolina
  - Family Medicine of Sayebrook, Myrtle Beach, South Carolina
  - Piedmont Research Partners, Old Point Station, South Carolina
  - Palmetto Research Center, LLC, Spartanburg, South Carolina
  - Palmetto Clinical Research, Summerville, South Carolina
  - PMG Research of Bristol, LLC, Bristol, Tennessee
  - Chattanooga Medical Research, LLC, Chattanooga, Tennessee
  - Chattanooga Research and Medicine (CHARM), Chattanooga, Tennessee
  - University Diabetes & Endocrine Consultants, Chattanooga, Tennessee
  - WR-ClinSearch, LLC, Chattanooga, Tennessee
  - Holston Medical Group, P.C., Kingsport, Tennessee
  - Metro Knoxville HMA, LLC, Knoxville, Tennessee
  - VA Medical Center - Memphis, Memphis, Tennessee
  - Tennessee Valley Healthcare System, Nashville, Tennessee
  - Central Texas Clinical Research, LLC, Austin, Texas
  - Protenium Clinical Research, Dallas, Texas
  - VA Medical Center - Dallas, Dallas, Texas
  - North Texas Endocrine Center, Dallas, Texas
  - Research Institute of Dallas, P.A., Dallas, Texas
  - Synexus Clinical Research US, Inc., Dallas, Texas
  - Doctors Hospital at Renaissance, Edinburg, Texas
  - Texas Health Research & Education Institute, Fort Worth, Texas
  - Texas Health Physicians Group, Fort Worth, Texas
  - University of North Texas Health Science Center, Fort Worth, Texas
  - Diabetes and Thyroid Center of Fort Worth, Fort Worth, Texas
  - Rockwood Medical Clinic, Fort Worth, Texas
  - East Texas Cardiology PA, Houston, Texas
  - Endocrine Associates, LLC, Houston, Texas
  - Heights Doctors Clinic, Houston, Texas
  - Associates in Medicine, Houston, Texas
  - Michael E. DeBakey VA Medical Center, Houston, Texas
  - Southwest Clinical Trials, Houston, Texas
  - Protenium Clinical Research, Hurst, Texas
  - Houston Methodist Research Institute - CCAT Pearland, Pearland, Texas
  - Clinical Investigations of Texas, Plano, Texas
  - Consano Clinical Research, LLC, San Antonio, Texas
  - Sant Antonio Premiere Internal Medicine, San Antonio, Texas
  - Briggs Clinical Research, LLC., San Antonio, Texas
  - Schnitzler Cardiovascular Consultants (SCC), PLLC, San Antonio, Texas
  - Bandera Family Healthcare Research LLC, San Antonio, Texas
  - Northeast Clinical Research of San Antonio, Schertz, Texas
  - Spring Family Practice Associates, Spring, Texas
  - Northwest Houston Heart Center, Tomball, Texas
  - Victoria Heart & Vascular Center, Victoria, Texas
  - Hillcrest Family Health Clinics, Waco, Texas
  - Utah Cardiology, P.C. (Davis), Farmington, Utah
  - VA Medical Center, White River Junction, Vermont
  - Burke Internal Medicine & Research, Burke, Virginia
  - Virginia Endocrinology Research, Chesapeake, Virginia
  - Carient Heart and Vascular, Manassas, Virginia
  - Clinical Research Partners, LLC, Richmond, Virginia
  - McGuire DVA Medical Center, Richmond, Virginia
  - Roanoke Heart Institute, Roanoke, Virginia
  - Suffolk Multispecialty Research, Suffolk, Virginia
  - Corporation Lane Internal Medicine, Virginia Beach, Virginia
  - Cardiology Associates of Bellin Health, Green Bay, Wisconsin
  - Clinical Investigation Specialists Inc, Kenosha, Wisconsin
  - Mayo Clinic Health System, La Crosse, Wisconsin
  - Meriter Medical Group, Inc., Madison, Wisconsin
  - Zablocki VA Medical Center, Milwaukee, Wisconsin
- Argentina (29):
  - Hospital Interzonal General de Agudos Dr Jose Penna, Bahía Blanca, Buenos Aires
  - Hospital Italiano Regional del Sur, Bahía Blanca, Buenos Aires
  - Hospital Italiano, Ciudad Autonoma Buenos Aires, Buenos Aires
  - CICLO, La Plata, Buenos Aires
  - Centro de Investigaciones Medicas Mar del Plata, Mar del Plata, Buenos Aires
  - Instituto de Investigaciones Clinicas, Mar del Plata, Buenos Aires
  - Instituto de Investigaciones Clinicas San Nicolas, San Nicolás de los Arroyos, Buenos Aires
  - Instituto Clinico Metabolico, San Nicolás de los Arroyos, Buenos Aires
  - Clinica Olivos, Vicente López, Buenos Aires
  - Centro Medico Viamonte SRL, Buenos Aires, Ciudad Autonoma Buenos Aires
  - Hospital Sirio Libanes, Caba, Ciudad Autonoma Buenos Aires
  - Sanatorio Güemes, Ciudad Autonoma de Bs. As., Ciudad Autonoma Buenos Aires
  - CEMEDIC - Centro de Especialidades Medicas, Villa Luro, Ciudad Autonoma Buenos Aires
  - Centro Medico Luquez, San Vicente, Córdoba Province
  - Axismed S.R.L.- Clínica Mayo, San Miguel de Tucumán, Tucumán Province
  - Consultorio Dr. Litvak Bruno, Ciudad Autonoma Buenos Aires
  - Fundacion Favaloro, Ciudad Autonoma Buenos Aires
  - CIPREC, Ciudad Autonoma Buenos Aires
  - Investigaciones Medicas IMOBA S.R.L, Ciudad Autonoma Buenos Aires
  - Centro Medico Dra Laura Maffei Investigacion Clinica Aplicada, Ciudad Autonoma Buenos Aires
  - CEDIC Centro de Investigaciones Clinicas, Ciudad Autonoma Buenos Aires
  - Instituto Cardiovascular Buenos Aires, Ciudad Autonoma Buenos Aires
  - CCBR - Buenos Aires - AR, Ciudad Autonoma Buenos Aires
  - Instituto de Cardiologia de Corrientes, Corrientes
  - Inst. Privado de Inv. Clinicas de Cordoba, Córdoba
  - Instituto Medico DAMIC, Córdoba
  - Hospital Privado Centro Medico de Cordoba S.A, Córdoba
  - Clinica del Prado, Córdoba
  - Prevencion Cardiovascular Salta, Salta
- Brazil (40):
  - L2IP - Instituto de Pesquisas Clínicas Ltda., Brasília, Federal District
  - Hospital do Coração do Brasil, Brasília, Federal District
  - CECAP - Centro de Cardiologia Clínica, Brasília, Federal District
  - Hospital Universitário de Brasília, Brasília, Federal District
  - Clínica de Endocrinologia e Metabologia Ltda., Brasília, Federal District
  - CARDIOINTERV Centro de Pesquisa S/S, Goiânia, Goiás
  - Via Médica, Goiânia, Goiás
  - HC-UFG - Hospital das Clínicas da Universidade Federal de Goiás, Goiânia, Goiás
  - Hospital Felício Rocho, Belo Horizonte, Minas Gerais
  - CARDRESEARCH - Cardiologia Assistencial, Belo Horizonte, Minas Gerais
  - Sociedade Hospitalar Angelina Caron, Campina Grande do Sul, Paraná
  - Cline Research Center (Leite PS Consultoria Medica LTDA), Curitiba, Paraná
  - Núcleo de Pesquisa Clínica S/S, Curitiba, Paraná
  - Paraná Medical Research Center, Maringá, Paraná
  - HUJBB-UFPA - Hospital Universitário João de Barros Barreto - Universidade Federal do Pará, Belém, Pará
  - CCBR Brasil Centro de Pesquisas e Análises Clínicas Ltda., Rio de Janeiro, Rio Do Janeiro
  - Eurolatino Natal Pesquisas Médicas Ltda., Natal, Rio Grande do Norte
  - Hospital Universitário, Canoas, Rio Grande do Sul
  - Hospital São Vicente de Paulo, Passo Fundo, Rio Grande do Sul
  - Santa Casa de Misericórdia de Pelotas, Pelotas, Rio Grande do Sul
  - Santa Casa de Misericórdia de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Centro de Pesquisas em Diabetes Ltda., Porto Alegre, Rio Grande do Sul
  - Centro de Pesquisa Clínica Maimônides - Maimônides Day Hospital, Porto Alegre, Rio Grande do Sul
  - Centro de Pesquisa Médica Santa Maria Ltda., Santa Maria, Rio Grande do Sul
  - Maestri e Kormann Consultoria Medico Científica LTDA, Blumenau, Santa Catarina
  - Loema - Instituto de Pesquisa Clínica, Campinas, São Paulo
  - IPCC - Instituto de Pesquisa Clínica de Campinas, Campinas, São Paulo
  - CEMEC - Centro Multidisciplinar de Estudos Clínicos, São Bernardo do Campo, São Paulo
  - Fundação Faculdade Regional de Medicina de São José do Rio Preto, São José do Rio Preto, São Paulo
  - ISPEM - Instituto São José dos Campos em Pesquisas Médicas, São José dos Campos, São Paulo
  - CPQuali Pesquisa Clínica Ltda., São Paulo, São Paulo
  - CPCLIN - Centro de Pesquisas Clínicas Ltda., São Paulo, São Paulo
  - Clínica Paulista de Doenças Cardiovasculares Ltda., São Paulo, São Paulo
  - Dr. Consulta, São Paulo, São Paulo
  - CEPIC - Centro Paulista de Investigação Clínica e Serviços Médicos, São Paulo, São Paulo
  - Hospital das Clínicas da Faculdade de Medicina da USP, São Paulo, São Paulo
  - Incor - Instituto do Coração - HCFMUSP, São Paulo, São Paulo
  - IMC - Instituto de Moléstias Cardiovasculares Tatuí, Tatuí, São Paulo
  - Santa Casa de Votuporanga, Votuporanga, São Paulo
- Bulgaria (32):
  - MHAT 'Puls' AD, Blagoevgrad
  - MHAT - Blagoevgrad, EOOD, Blagoevgrad
  - MHAT "Yuliya Vrevska - Byala", EOOD, Byala
  - MHAT-Haskovo, AD, Haskovo
  - MHAT "Higia", AD - Pazardzhik, Pazardzhik
  - MHAT - Pazardzhik AD, Pazardzhik
  - MHAT "Sv. Pantaleymon - Pleven", OOD, Pleven
  - SHATC Pleven EAD, Pleven
  - UMHAT 'Dr. Georgi Stranski', EAD, Pleven
  - UMHAT "Sv. Georgi", EAD, Plovdiv
  - UMHAT "Kaspela", EOOD, Plovdiv
  - MC Rusemed ltd., Rousse
  - Diagnostic Consultative Center II - Sofia OOD, Sofia
  - Fifth MHAT - Sofia EAD, Sofia
  - NMTH "Tsar Boris III", Sofia
  - MHAT - "National Heart Hospital" EAD, Sofia
  - MHAT "Lyulin", EAD, Sofia
  - Acibadem City Clinic Tokuda Hospital Ead, Sofia
  - MC Start - d-r Todor Dimitrov EOOD, Sofia
  - DCC "Alexandrovska", EOOD, Sofia
  - UMHAT "Alexandrovska" EAD, Sofia
  - UMHAT 'Tsaritsa Yoanna - ISUL', EAD, Sofia
  - Fourth MHAT - Sofia EAD, Sofia
  - Diagnostic Consultation Center CONVEX EOOD, Sofia
  - Medical Center Kalimat, Sofia
  - UMHAT 'Sveta Anna' AD, Sofia
  - MC "Synexus - Sofia", EOOD, Sofia
  - UMHAT "SofiaMed", OOD, Sofia
  - MC "Orfey", EOOD, Stara Zagora
  - SHATC "Cardiolife", OOD, Varna
  - SHATC - Varna, EOOD, Varna
  - MHAT "Sv. Panteleymon", AD, Yambol
- Canada (51):
  - LMC Clinical Research Inc. (Calgary), Calgary, Alberta
  - ALTA Clinical Research Inc., Edmonton, Alberta
  - Royal Alexandra Hospital, CK Hui Heart Centre, Edmonton, Alberta
  - The Bailey Clinic, Red Deer, Alberta
  - Fraser Clinical Trials Inc., New Westminster, British Columbia
  - Surrey Memorial Hospital, Surrey, British Columbia
  - BC Diabetes As Operated by Dr. TG Elliott, Inc., Vancouver, British Columbia
  - Discovery Clinical Services Ltd., Victoria, British Columbia
  - Saint Boniface General Hospital, Winnipeg, Manitoba
  - Rivergrove Medical Clinic, Winnipeg, Manitoba
  - Winnipeg Clinic, Winnipeg, Manitoba
  - Health Sciences Centre, St. John's, Newfoundland and Labrador
  - LMC Clinical Research Inc. (Barrie), Barrie, Ontario
  - LMC Clinical Research Inc. (Brampton), Brampton, Ontario
  - Aggarwal and Associates Ltd, Brampton, Ontario
  - JBN Medical Diagnostic Services Inc., Burlington, Ontario
  - LMC Clinical Research dba Manna Research Inc. Burlington North, Burlington, Ontario
  - Cambridge Cardiac Care Centre, Cambridge, Ontario
  - Joanne F. Liutkus Medicine Professional Corporation, Cambridge, Ontario
  - Saul Vizel Professional Medicine Corporation, Cambridge, Ontario
  - LMC Clinical Research Inc. (Thornhill), Concord, Ontario
  - LMC Clinical Research Inc. (Etobicoke), Etobicoke, Ontario
  - Janik Research, Greater Sudbury, Ontario
  - Dawson Road Family Medical Clinic, Guelph, Ontario
  - LMC Clinical Research Inc. (Ottawa), Nepean, Ontario
  - LMC Clinical Research Inc. (Oakville), Oakville, Ontario
  - James Cha, MD, Oshawa, Ontario
  - The Ottawa Hospital - Riverside Campus, Ottawa, Ontario
  - Kawartha Cardiology Clinical Trials, Peterborough, Ontario
  - Scarborough Cardiology Research, Scarborough Village, Ontario
  - Humber River Hospital, Toronto, Ontario
  - LMC Clinical Research Inc. (Bayview), Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - LMC Clinical Research dba Manna Research Inc. Toronto, Toronto, Ontario
  - Ecogene-21, Chicoutimi, Quebec
  - ViaCar Recherche Clinique Inc, Greenfield Park, Quebec
  - Clinique de Cardiologie de Levis, Lévis, Quebec
  - Centre de Dépistage et Recherche Cardiovasculaire Rive-Sud, Longueuil, Quebec
  - LMC Clinical Research dba Manna Research Inc. Mirabel, Mirabel, Quebec
  - Clinique Santé Cardio MC, Montreal, Quebec
  - CHUM Hôtel-Dieu, Montreal, Quebec
  - Applied Medical Informatics Research Inc., Montreal, Quebec
  - Recherche Clinique Sigma Inc., Québec, Quebec
  - Clinique Médicale St-Louis (Recherche) inc d/b/a/ Centre de Recherche Saint-Louis, Québec, Quebec
  - ALPHA Recherche Clinique, Québec, Quebec
  - Recherche Médicale St-Jérôme Inc., Saint-Jérôme, Quebec
  - LMC Clinical Research Inc. (Montreal), Saint-Laurent, Quebec
  - Centre Medical des Carrieres, Saint-Marc-des-Carrieres, Quebec
  - DIEX Recherche Quebec Inc., Québec
  - Institut Universitaire de Cardiologie et de Pneumologie de Quebec, Québec
  - Clinique des maladies Lipidiques de Quebec, Québec
- Colombia (8):
  - Centro de Investigacion Medico Asistencial S.A.S, Barranquilla
  - IPS Centro Cientifico Asistencial S.A.S, Barranquilla
  - Dexa Diab Servicios Médicos Limitada., Bogotá
  - Solano y Terront Servicios Médicos Ltda., Bogotá
  - Centro Cardiovascular Aristides Sotomayor Santa Lucia S.A.S. - IPS ASTALUC S.A.S. IPS, Cartagena
  - Fundación Centro de Investigaciones Biomédicas Riescard, Espinal
  - Fundación Oftalmológica de Santander - FOSCAL, Floridablanca
  - Centro de Investigación Clínica CIC, Medellín
- Czechia (26):
  - Medicentrum Beroun spol. s.r.o., Beroun
  - Nemocnice Milosrdnych bratri, Brno
  - Fakultni nemocnice u sv. Anny v Brne, Brno
  - EDUMED s.r.o, Broumov
  - Poliklinika Chocen a.s., Choceň
  - Ordinace pro choroby srdce s.r.o., Chomutov
  - MUDr. Jan Hubac s.r.o., Chrudim
  - Nemocnice Havlickuv Brod p.o., Havlíčkův Brod
  - Kardio-Pisova s.r.o., Hradec Králové
  - MUDr. Tomas Edelsberger, Krnov
  - EDUMED s.r.o, Náchod
  - Agentura Science Pro Spol. s.r.o., Olomouc
  - PreventaMed s.r.o., Olomouc
  - CCR Ostrava s.r.o., Ostrava
  - MUDr. Jan KVASNICKA CSc. Angiologie kardiologie a interna, Prague
  - Nemocnice na Frantisku, Prague
  - Synexus Czech s.r.o., Prague
  - Vseobecna fakultni nemocnice v Praze, Prague
  - Corintez s.r.o., Prague
  - ResTrial s.r.o., Prague
  - MUDr.Eva Mandakova MBA, Rakovník
  - Nemocnice Slany, Slaný
  - AeskuLab k.s., Teplice
  - Kardiologicka ambulance MUDr. Ferkl s.r.o., Trutnov
  - Clinical Trials Services s.r.o, Uherské Hradiště
  - MUDr. Nina Zemkova s.r.o., Uherské Hradiště
- Denmark (14):
  - Bioclinica, Aalborg
  - Ålborg Universitets Hospital, Aalborg
  - Aarhus University Hospital, Aarhus
  - Bioclinica, Ballerup Municipality
  - Amager-Hvidovre Hospital, Copenhagen S
  - Sydvestjyds Sygehus Esbjerg, Esbjerg
  - Amager-Hvidovre Hospital, Glostrup Municipality
  - Herlev og Gentofte Hospital, Hellerup
  - Herlev og Gentofte Hospital, Herlev
  - Regionshospitalet Herning-Hospitalsenheden Vest, Herning
  - Holbæk Sygehus, Holbæk
  - Sjællands Universitetshospital, Roskilde
  - OUH, Svendborg
  - Bioclinica, Vejle
- France (3):
  - CHU Tours - Hôpital Trousseau, Chambray-lès-Tours, Indre Et Loire
  - CHU Nantes - Hopital Nord Laënnec, Nantes, Loire Atlantique
  - Hôpital Bichat - Claude Bernard, Paris, Paris
- Germany (27):
  - Universitaetsklinikum Freiburg, Freiburg im Breisgau, Baden-Wurttemberg
  - Praxis fuer Praevention und Therapie, Villingen-Schwenningen, Baden-Wurttemberg
  - Gemeinschaftspraxis Dr. Klein/ Minnich, Künzing, Bavaria
  - Klinikum der Universitaet Muenchen, Munich, Bavaria
  - Deutsches Herzzentrum Muenchen, Munich, Bavaria
  - GP Dr. Haggenmiller, PD Dr. Michael Jeserich, Naumburg, Bavaria
  - ZKS-Südbrandenburg -center for clinical studies Südbrandenburg GmbH, Elsterwerda, Brandenburg
  - Neurologische Praxis Dr. Schoell & Kollegen, Bad Homburg, Hesse
  - Synexus Clinical Research GmbH, Frankfurt am Main, Hesse
  - ClinPhenomics GmbH & Co KG, Frankfurt am Main, Hesse
  - Klinische Forschung Schwerin GmbH, Schwerin, Mecklenburg-Vorpommern
  - Synexus Clinical Research GmbH, Bochum, North Rhine-Westphalia
  - Gemeinschaftspraxis Diabeteszentrum Dortmund Dr.med. Klaus Busch, Dortmund, North Rhine-Westphalia
  - Kardiologische Praxis Gemeinschaftspraxis, Dortmund, North Rhine-Westphalia
  - St. Johannes Hospital, Dortmund, North Rhine-Westphalia
  - Klinikum Bielefeld gem. GmbH, Dortmund, North Rhine-Westphalia
  - Zentrum fuer Praevention und Rehabilitation, Siegen, North Rhine-Westphalia
  - Synexus Clinical Research GmbH, Leipzig, Saxony
  - Gemeinschaftspraxis Dr. Taeschner / Dr. Bonigut, Leipzig, Saxony
  - Dr. Uwe Böckmann / Birgit Jacobs - Diabeteszentrum Neumünster, Neumünster, Schleswig-Holstein
  - RED - Institut GmbH, Oldenburg in Holstein, Schleswig-Holstein
  - Katholisches Krankenhaus "St. Johann Nepomuk", Erfurt, Thuringia
  - Diabetespraxis Prenzlauer Allee, Berlin
  - Institut fuer klinische Forschung und Entwicklung Berlin GmbH, Berlin
  - Studienzentrum Rankestrasse, Berlin
  - Synexus Clinical Research GmbH, Berlin
  - Gemeinschaftspraxis fuer innere Medizin und Diabetologie, Hamburg
- Hungary (28):
  - Lausmed Kft., Baja
  - Principal SMO Kft., Baja
  - DRC Gyogyszervizsgalo Kozpont Kft., Balatonfüred
  - Bekes Megyei Kozponti Korhaz Dr. Rethy Pal Tagkorhaz, Békéscsaba
  - Belgyogyaszati es Kardiologiai Maganrendelo, Békéscsaba
  - Clinexpert Kft., Budapest
  - Synexus Magyarorszag Kft., Budapest
  - CSALADGYOGYASZ Kft., Budapest
  - Semmelweis Egyetem, Budapest
  - Borvo Clinic Kft., Debrecen
  - Debreceni Egyetem, Debrecen
  - Meditoll Kft., Gödöllő
  - Bekes Megyei Kozponti Korhaz Pandy Kalman Tagkorhaza, Gyula
  - Synexus Magyarorszag Egeszsegugyi Szolgaltato Kft.- Gyula DRS, Gyula
  - BKS Research Kft., Hatvan
  - Z+P MED Egeszsegugyi, Kereskedelmi es Szolgaltato Bt., Kalocsa
  - Somogy Megyei Kaposi Mor Oktato Korhaz, Kaposvár
  - Selye Janos Korhaz, Komárom
  - IPR Hungary Kft., Miskolc
  - Kanizsai Dorottya Korhaz, Nagykanizsa
  - Medifarma-98 Kft., Nyíregyháza
  - BORBANYA PRAXIS Kft., Nyíregyháza
  - Dr. Nagy Laszlo Kardiologiai Maganrendeles, Orosháza
  - Da Vinci Maganklinika, Pécs
  - Tolna Megyei Balassa Janos Korhaz, Szekszárd
  - Fejer Megyei Szent Gyorgy Egyetemi Oktato Korhaz, Székesfehérvár
  - Csolnoky Ferenc Korhaz, Veszprém
  - Zala Megyei Szent Rafael Korhaz, Zalaegerszeg
- India (31):
  - Vijaya Super Speciality Hospital, Nellore, Andhra Pradesh
  - GNRC Hospital, Guwahati, Assam
  - Ahmedabad Bariatrics and Cosmetics Pvt Ltd., Ahmedabad, Gujarat
  - S. A. L. Hospital & Medical Institute, Ahmedabad, Gujarat
  - DDMM Heart Institute, Nadiād, Gujarat
  - Shri B. D. Mehta Mahavir Heart Institute, Surat, Gujarat
  - BAPS Pramukhswami Hospital, Surat, Gujarat
  - Sterling Hospital, Vadodara, Gujarat
  - Rhythm Heart Institute, Vadodara, Gujarat
  - Medanta The Medicity, Gurgaon, Haryana
  - Fortis Hospitals Ltd., Bangalore, Karnataka
  - K.L.E. Society's Dr. Prabhakar Kore Hospital and Medical Research Centre, Belagavi, Karnataka
  - JSS Hospital, Mysuru, Karnataka
  - Medical College, Thiruvananthapuram, Kerala
  - Meditrina Institute Of Medical Sciences, Nagpur, Maharashtra
  - Supe Heart & Diabetes Hospital & Research Centre, Nashik, Maharashtra
  - 7-Orange Hospital, Pimpri-Chinchwad, Maharashtra
  - Shree Multispecialty Hospital, Pune, Maharashtra
  - King Edward Memorial Hospital Research Centre, Pune, Maharashtra
  - Aashirwad Hospital, Ulhasnagar, Maharashtra
  - Loknayak Hospital, New Delhi, National Capital Territory of Delhi
  - Sir Gangaram Hospital, New Delhi, National Capital Territory of Delhi
  - Fortis Flight Lieutenant Rajan Dhall Hospital, New Delhi, National Capital Territory of Delhi
  - Institute of Medical Sciences and SUM Hospital, Bhubaneshwar, Odisha
  - Eternal Heart Care Centre, Jaipur, Rajasthan
  - SRM Institutes for Medical Sciences, Chennai, Tamil Nadu
  - Institute of Cardiovascular Diseases Madras Medical Mission, Chennai, Tamil Nadu
  - KRM Hospital & Research Centre, Lucknow, Uttar Pradesh
  - Galaxy Hospital, Varanasi, Uttar Pradesh
  - IPGMER and SSKM Hospital, Kolkata, West Bengal
  - Maharaja Agrasen Hospital, Delhi
- Israel (14):
  - HaEmek Medical Center, Afula
  - Bnai Zion Medical Center, Haifa
  - Rambam Health Care Center, Haifa
  - The Lady Davis Carmel Medical Center, Haifa
  - Wolfson Medical Center, Holon
  - Shaare Zedek Medical Center, Jerusalem
  - Hadassah University Hospital - Ein Kerem, Jerusalem
  - Galilee Medical Center, Nahariya
  - Rabin Medical Center-Beilinson Campus, Petah Tikva
  - Chaim Sheba Medical Center, Ramat Gan
  - Kaplan Medical Center, Rehovot
  - Ziv Medical Center, Safed
  - Tel Aviv Sourasky Medical Center, Tel Aviv
  - Diabetes Medical Center, Tel Aviv
- Japan (64):
  - Aichi Medical University Hospital, Nagakute-shi, Aichi-ken
  - JOHAS Chubu Rosai Hospital, Nagoya, Aichi-ken
  - Kojunkai Daido Clinic, Nagoya, Aichi-ken
  - NHO Nagoya Medical Center, Nagoya, Aichi-ken
  - National Center For Geriatrics And Gerontology, Obu-shi, Aichi-ken
  - Fujita Health University Hospital, Toyoake-shi, Aichi-ken
  - Chiba University Hospital, Chiba, Chiba
  - Kioroshikai Chibanishi General Hospital, Matsudo-shi, Chiba
  - Seikeikai New Tokyo Heart Clinic, Matsudo-shi, Chiba
  - Ehime Prefectural Central Hospital, Matsuyama, Ehime
  - Fukuoka University Hospital, Fukuoka, Fukuoka
  - Fukuoka Tokushukai Hospital, Kasuga-shi, Fukuoka
  - Steel Memorial Yawata Hospital, Kitakyushu-shi, Fukuoka
  - NHO Fukuoka Higashi Medical Center, Koga-shi, Fukuoka
  - Chiyukai Fukuoka Shinmizumaki Hospital, Onga-gun, Fukuoka
  - Southern Tohoku Medical Clinic, Koriyama-shi, Fukushima
  - Hoshi General Hospital, Koriyama-shi, Fukushima
  - Nakahama Heart Clinic, Fuchu-shi, Hiroshima
  - Nippon Kokan Fukuyama Hospital, Fukuyama-shi, Hiroshima
  - NHO Higashihiroshima Medical Center, Higashihiroshima-shi, Hiroshima
  - Miyanosawa Clinic of Internal Medicine and Cardiology, Sapporo, Hokkaido
  - Tanaka Cardiology Clinic, Hitachi-Naka, Ibaraki
  - Nakakinen Clinic Medical Corporation Kensei-kai, Naka, Ibaraki
  - Public Central Hospital of Matto Ishikawa, Hakusan-shi, Ishikawa-ken
  - NHI Komatsu Municipal Hospital, Komatsu-shi, Ishikawa-ken
  - Kuonkai Kamata Medical Clinic, Morioka, Iwate
  - Iwate Medical University Uchimaru Medical Center Hospital, Morioka, Iwate
  - Josuikai Olive Takamatsu Medical Clinic, Takamatsu, Kagawa-ken
  - Sohken Yamamoto Clinic, Sagamihara-shi, Kanagawa
  - NHO Yokohama Medical Center, Yokohama, Kanagawa
  - Kumamoto University Hospital, Kumamoto, Kumamoto
  - Ryubokai Higashi Diabetes and Cardiovascular Clinic, Tamana-shi, Kumamoto
  - Ijinkai Takeda General Hospital, Kyoto, Kyoto
  - Kyoto University Hospital, Kyoto, Kyoto
  - Rakuwakai Otowa Hospital, Kyoto, Kyoto
  - Sato Hospital, Osaki-shi, Miyagi
  - Tohoku Kosai Hospital, Sendai, Miyagi
  - Sendai Kousei Hospital, Sendai, Miyagi
  - Keiwakai Oita Oka Hospital, Ōita, Oita Prefecture
  - Okayama University Hospital, Okayama, Okayama-ken
  - Okinawa Tokushukai Chubu Tokushukai Hospital, Nakagami-gun, Okinawa
  - Iwasaki Naika Clinic, Higashiosaka-shi, Osaka
  - Takekawa Naika Clinic, Higashiosaka-shi, Osaka
  - Rinku General Medical Center, Izumisano, Osaka
  - Shiraiwa Medical Clinic, Kashiwara-shi, Osaka
  - Tokushukai Kishiwada Tokushukai Hospital, Kishiwada-shi, Osaka
  - Kansai Electric Power Hospital, Osaka, Osaka
  - National Cerebral and Cardiovascular Center, Suita-shi, Osaka
  - Senrichuo Ekimae Clinic, Toyonaka-shi, Osaka
  - IMS Miyoshi General Hospital, Iruma-gun, Saitama
  - Sugiura Clinic, Kawaguchi-shi, Saitama
  - Sanyukai Saino Clinic, Tokorozawa-shi, Saitama
  - NHO Saitama National Hospital, Wako-shi, Saitama
  - Shiga University of Medical Science Hospital, Ōtsu, Shiga
  - NHO Hamada Medical Center, Hamada-shi, Shimane
  - Jichi Medical University Hospital, Shimotsuke-shi, Tochigi
  - Juntendo University Hospital, Bunkyō City, Tokyo-To
  - Fukuwa Clinic, Chūōku, Tokyo-To
  - Tokyo-Eki Center-Building Clinic, Chūōku, Tokyo-To
  - Nomura Clinic, Itabashi-ku, Tokyo-To
  - Hosoda Clinic, Katsushika-ku, Tokyo-To
  - Toyukai Yutenji Medical Clinic (Yutenji Naika), Meguro-ku, Tokyo-To
  - Shinjuku Research Park Clinic, Shinjuku-ku, Tokyo-To
  - Yamaguchi University Hospital, Ube-shi, Yamaguchi
- Mexico (18):
  - Centro de Investigacion Cardiovascular y Metabolica, Tijuana, Baja California Norte
  - Centro de Investigacion Clinica del Pacifico, S.A. de C.V., Acapulco de Juárez, Guerrero
  - Cardiologia Clinica e Intervencionista, Guadalajara, Jalisco
  - Centro de Investigacion Medica de Occidente, S.C., Zapopan, Jalisco
  - Phytomedicamenta S.A. de C.V., Mexico City, Mexico City
  - Health Pharma Professional Research S.A. de C.V., Mexico City, Mexico City
  - Centro de Atención e Investigación en Factores de Riesgo Cardiovascular Omega S.C., Mexico City, Mexico City
  - Instituto Nacional de Ciencias Médicas y Nutricion Dr. Salvador Zubiran, Mexico City, Mexico City
  - Mentrials S.A. de C.V., Mexico City, Mexico City
  - Instituto de Diabetes, Obesidad y Nutrición S.C., Cuautla, Morelos
  - Universidad Autonoma de Nuevo Leon, Hospital Universitario Dr. Jose Eleuterio Gonzalez, Monterrey, Nuevo León
  - Centro Medico San Francisco, Monterrey, Nuevo León
  - Unidad Medica para la Salud Integral, San Nicolás de los Garza, Nuevo León
  - Centro Integral Medico SJR S.C., San Juan del Río, Querétaro
  - Centro de Estudios de Investigacion Metabolicos y Cardiovasculares S.C., Madero, Tamaulipas
  - Centro de Investigacion Cardiometabolica de Aguascalientes S.A de C.V, Aguascalientes
  - Investigacion En Salud Y Metabolismo S.C., Chihuahua City
  - Sociedad de Metabolismo y Corazon S.C, Veracruz
- Netherlands (27):
  - Noordwest Ziekenhuisgroep, Alkmaar
  - Ziekenhuisgroep Twente, Almelo, Almelo
  - Meander Medisch Centrum, Amersfoort
  - Ziekenhuis Amstelland, Amstelveen
  - BovenlJ Ziekenhuis, Amsterdam
  - Amsterdam UMC, Locatie AMC, Amsterdam
  - Gelre ziekenhuizen, locatie Lukas, Apeldoorn
  - Rijnstate, Arnhem
  - Deventer Ziekenhuis, Deventer
  - Albert Schweitzer Ziekenhuis, Dordwijk, Dordrecht
  - Gelderse Vallei Ziekenhuis, Ede, Ede
  - Catharina Ziekenhuis Eindhoven, Eindhoven
  - Spaarne Gasthuis, Hoofddorp, Haarlem
  - Zuyderland Medisch Centrum - Heerlen, Heerlen
  - Huisartsenpraktijk Gorecht, Hoogezand
  - Quality Care Research, Kloosterhaar
  - Leids Universitair Medisch Centrum, Leiden
  - Bravis Ziekenhuis, Roosendaal, Roosendaal
  - Maasstad Ziekenhuis, Zuider, Rotterdam
  - Ikazia Ziekenhuis, Rotterdam
  - Albert Schweitzer Ziekenhuis, Zwijndrecht, Sliedrecht
  - Haga Ziekenhuis, The Hague
  - Bernhoven Uden, Uden
  - UMC Utrecht, Utrecht
  - Diakonessenhuis, Utrecht, Utrecht
  - Maxima Medisch Centrum, Veldhoven
  - VieCuri Medisch Centrum, Venlo
- Poland (38):
  - NZOZ Centrum Medyczne KERmed, Bydgoszcz
  - KARDIOMED Janczska Kociwska Ostki PodckaRekrzSp, Elblag
  - Poradnia Kardiologiczna Jarosław Jurowiecki, Gdansk
  - Synexus Polska SCM Sp. z o.o. Gdansku, Gdansk
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Indywidualna Specjalistyczna Praktyka Lekarska w Dziedzinie Kardiologii lek. med. Krzysztof Cymerman, Gdynia
  - Synexus Polska Sp. z o.o. Oddzial w Gdyni, Gdynia
  - Samodzielny Publiczny Specjalistyczny Szpital Zachodni im. Jana Pawla II, Grodzisk Mazowiecki
  - Synexus Polska Sp. z o.o. Oddzial w Katowicach, Katowice
  - Centrum Medyczne Pratia Katowice II, Katowice
  - SPSK Nr 7 SUM w Katowicach Gornoslaskie CM im. prof. Leszka Gieca, Katowice
  - Specjalistyczna Poradnia Kardiologiczna i Nadciśnienia Tętniczego, Kielce
  - Augustyn Monika, Krakow
  - Krakowskie Centrum Medyczne Sp. z o.o., Krakow
  - Wojewódzkie Wielospecjalistyczne Centrum Onkologii i Traumatologii im. M. Kopernika w Łodzi, Lodz
  - NZOZ ALL-MED Centrum Medyczne Specjalistyczne Gabinety Lekarskie, Lodz
  - Indywidualna Specjalistyczna Praktyka Lekarska, Lodz
  - KO-MED Centra Kliniczne Lublin II, Lublin
  - Clinical Best Solutions, Lublin
  - NZOZ Twoja Przychodnia, Lublin
  - NZOZ Osrodek Kardiologii Inwazyjnej -Ikardia, Nałęczów
  - Medicome Sp. z o.o., Oświęcim
  - Synexus Polska sp. z o.o. Oddzial w Poznaniu, Poznan
  - Praktyka Lekarska Ewa Krzyzagorska, Poznan
  - KO-MED Centra Kliniczne Pulawy, Puławy
  - NZOZ Przychodnia Specjalistyczna H. Rudzki, A. Wittek, Ruda Śląska
  - Centrum Medyczne Medyk, Rzeszów
  - Clinmed Research, Skierniewice
  - NZOZ Pro-Cordis Sopockie Centrum Bad. Kardiolog., Sopot
  - KO-MED Centra Kliniczne Staszow, Staszów
  - Indywidualna Specjalistyczna Praktyka Lekarska dr n. med. Agnieszka Karczmarczyk Specjalista Chorob, Szczecin
  - NSZOZ Medicus, Środa Wielkopolska
  - NBR Polska, Warsaw
  - Centrum Medyczne Świat Pacjenta, Warsaw
  - Synexus Polska Sp. z o.o. Oddział w Warszawie, Warsaw
  - Centrum Zdrowia Tuchow Sp. z o.o., Wierzchosławice
  - Synexus Polska Sp. z o.o. Oddział we Wroclawiu, Wroclaw
  - KO-MED Centra Kliniczne Zamosc, Zamość
- VA Medical Center - San Juan, San Juan, Puerto Rico
- Romania (19):
  - S.C. CMI Dr. Pletea Noemi S.R.L, Bacau
  - Cabinet Medical Individual Diabet, Nutritie, Boli Metabolice Dr. Pop Lavinia, Baia Mare
  - S.C Centrul Medical de Diagnostic si Tratament Ambulator Neomed S.R.L, Brasov
  - S.C Clinica Medicala Data Plus S.R.L, Bucharest
  - Spitalul Clinic Colentina, Bucharest
  - Spitalul Clinic de Urgenta "Sfantul Pantelimon", Bucharest
  - Institutul de Urgenta pentru Boli Cardiovasculare "Prof. Dr. C.C. Iliescu", Bucharest
  - S.C. Health Net S.R.L, Bucharest
  - S.C Policlinica CCBR S.R.L, Bucharest
  - CMI Dr. Stolea T. Violeta - Medic specialist diabet zaharat, nutritie si boli metabolice, Bucharest
  - S.C. Medcon S.R.L., Buzău
  - S.C Grandmed S.R.L, Oradea
  - S.C Pelican Impex S.R.L, Oradea
  - S.C. Bella Praxis S.R.L, Pașcani
  - S.C. Diabmed Dr. Popescu Alexandrina S.R.L, Ploieşti
  - CMI Dr Busegeanu Mihaela Magdalena, Ploieşti
  - S.C Mediab S.R.L, Târgu Mureş
  - S.C Medicali's S.R.L, Timișoara
  - Spitalul Clinic Judetean de Urgenta "Pius Brinzeu", Timișoara
- Russia (40):
  - SBIH of Arkhangelsk region " First City Clinical hospital n.a. E. E. Volosevich", Arkhangelsk
  - TSHI "Altay Territorial Cardiologocal dispensary", Barnaul
  - FSHI "MSU of MoIA of RF of Kemerovo Region", Kemerovo
  - FSBI "Scientific-research Institute for Complex Problems of cardiovascular disease", Kemerovo
  - NSIH "Departmental Hospital on Station Kemerovo of OJSC "Russian Railways", Kemerovo
  - SAIH "Kemerovo Regional Clinical Hospital", Kemerovo
  - TSBIH "Krasnoyarsk Interdistrict Clinical Hospital of Emergency Medical Care n.a. N.S. Karpovich, Krasnoyarsk
  - SBIH of Moscow "City Clinical Hospital n.a.Bakhrushinykh", Moscow
  - SBHI "City Polyclinic #2 of Healthcare department of city of Moscow", Moscow
  - FSBIH "Central Clinical Hospital of Russian Academy of Sciences", Moscow
  - FSBI "Central Clinical Hospital with Polyclinic of the Department for Presidential Affairs of the RF, Moscow
  - SBEI HPE "Moscow State Medical and Dentistry University n.a. A. I. Evdokimov" of the MoH of the RF, Moscow
  - Murmansk Regional Clinical Hospital named after Bayandin, Murmansk
  - SBIH of Novosibirsk Region "Clinical Emergency Hospital #2", Novosibirsk
  - SBIH of Novosibirsk region "City Clinical Hospital # 19", Novosibirsk
  - FSBSI "Scientific Research Institute of Therapy and Preventive Medicine", Novosibirsk
  - LLC "RC Medical", Novosibirsk
  - BIH of Omsk region "Clinical Medico-Sanitary Unit # 9, Omsk
  - Llc Ultramed, Omsk
  - SBIH of Perm territory " City Clinical Hospital # 2 n.a. Fedor Khristoforovich Gral", Perm
  - State Budgetary Healthcare Institution Clinical Medical Sani, Perm
  - SHI "Perm Regional Hospital of War Veterans", Perm
  - City Emergency Hospital #2, Rostov-on-Don
  - CJSC Clinic complex, Saint Petersburg
  - FSBI North-West Federal Medical Research Center n.a. V.A. Almazov of MoH RF, Saint Petersburg
  - SPb SBIH "City Multy-field Hospital # 2", Saint Petersburg
  - Saint-Petersburg SBHI "City outpatient clinic #28", Saint Petersburg
  - LLC "Institute of Medical Examinations", Saint Petersburg
  - Pavlov First Saint Petersburg State Medical University, Saint Petersburg
  - Llc "Medinet", Saint Petersburg
  - SPb SBIH "Nikolaevskaya Hospital", Saint Petersburg
  - SPb SBIH "City Pokrovskaya Hospital", Saint Petersburg
  - LLC Medical Center Mart, Saint Petersburg
  - SIH "Saratov City Clinical Hospital # 2 n.a. V.I. Razumovskiy", Saratov
  - SPb SBIH "City Hospital # 40 of Kurortnyi region", Sestroretsk
  - FSBI "Research Institute for Cardiology" of Siberian Branch RAMS, Tomsk
  - SHI "Regional Clinical Hospital", Tver'
  - SHI Ulyanovsk Reg Clinical Hospital, Ulyanovsk
  - Yaroslavl Regional Clinical Hospital of War Veterans, Yaroslavl
  - SEIHPE "Ural SMA of RosZdrav" b.o. LLC "City Hospital #41", Yekaterinburg
- Slovakia (29):
  - Alian s.r.o., Bardejov
  - Thyreomedical s.r.o., Bardejov
  - Metabol KLINIK s.r.o., Bratislava
  - Galenum, s.r.o., Bratislava
  - DIAFA s.r.o., Bratislava
  - Diabet, spol. s.r.o., Bratislava
  - Kardiovaskularne centrum, s.r.o., Bratislava
  - Kardiologicka, interna a sonograficka amb. Kardio-Sanus, sro, Bratislava
  - MEDISPEKTRUM PLUS s.r.o., Bratislava
  - MUDr. Vladimir Gergel, s.r.o., Bratislava
  - ENDIAMED, s.r.o., Dolný Kubín
  - MEDICUS plus s.r.o., Komárno
  - Human-Care s.r.o., Košice
  - Sukromna interna a kardiologicka ambulancia, Košice
  - DIA- Kontrol s.r.o., Levice
  - CELL B, s.r.o., Levice
  - KARDIO 1 s.r.o., Lučenec
  - IN-DIA s.r.o., Lučenec
  - MUDr. Zuzana Ochodnicka,, Nitra
  - Fakultna nemocnica s poliklinikou Nove Zamky, Nové Zámky
  - DIABETOL s.r.o., Prešov
  - Medispol s.r.o., Prešov
  - Nemocnica s poliklinikou sv. Barbory Roznava a.s., Rožňava
  - Interna SK s.r.o., Svidník
  - Nemocnica arm. generala L. Svobodu Svidnik, a.s.,, Svidník
  - Peter Farkas MD, s.r.o., Šahy
  - Diabetes centrum, s.r.o., Trenčín
  - JAL s.r.o., Trnava
  - MEDIVASA s.r.o., Žilina
- South Africa (22):
  - Cardiology Clinical Research, Alberton, Gauteng
  - Johese Clinical Research: Unitas, Centurion, Gauteng
  - Medicross Roodepoort Clinical Research, Johannesburg, Gauteng
  - Lenasia Clinical Trial Centre, Johannesburg, Gauteng
  - Wits Clinical Research, Johannesburg, Gauteng
  - Clinresco Centres (Pty) Ltd, Kempton Park, Gauteng
  - Synexus SA - Stanza Clinical Research Centre, Mamelodi East, Gauteng
  - Seeber, M, Pretoria, Gauteng
  - Emmed Research, Pretoria, Gauteng
  - Synexus SA Watermeyer Clinical Research Centre, Pretoria, Gauteng
  - Johese Clinical Research: Midstream, Pretoria, Gauteng
  - Limpopo Clinical Research Initiative, Thabazimbi, Limpopo
  - Dr AA Mahomed Medical Centre, Moloto South, Mpumalanga
  - Synexus Helderberg Clinical Research Centre, Cape Town, Western Cape
  - Corbod Research, Cape Town, Western Cape
  - Tread Research, Cape Town, Western Cape
  - Tiervlei Trial Centre, Cape Town, Western Cape
  - Cape Town Medical Research Centre, Cape Town, Western Cape
  - Paarl Research Centre, Cape Town, Western Cape
  - Groote Schuur Hospital Lipid Laboratory, Cape Town, Western Cape
  - Dr JM Engelbrecht Practice, Somerset West, Western Cape
  - Helderberg Research Institute, Somerset West, Western Cape
- Spain (15):
  - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Virgen del Camino, Sanlúcar de Barrameda, Cádiz
  - Hospital Universitario Reina Sofia, Córdoba, Córdoba
  - Complejo Hospitalario Universitario A Coruña, A Coruña, La Coruña
  - Complejo Hospitalario Universitario de Santiago, Santiago de Compostela, La Coruña
  - Hospital Virgen del Mar, Almería
  - Hospital del Mar, Barcelona
  - Hospital Quironsalud Barcelona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Regional Universitario de Malaga, Málaga
  - Nuevas tecnologías en Diabetes y Endocrinología, Seville
  - Hospital Quironsalud Infanta Luisa, Seville
  - Hospital Universitario Virgen Macarena, Seville
- Ukraine (48):
  - Cherkasy Regional Cardiological Center, Cherkasy
  - CI Cherkasy RH of Cherkasy Regional Council, Cherkasy
  - CMI CCH#3 Dep of Ther# w the beds of card profile HSEI of UBSMU, Chernivtsi
  - RCI Chernivtsi Regional Endocrinology Center Policlinic Dept SHEI of UBSMU, Chernivtsi
  - CI Dnipropetrovsk City Cl Hosp #9 of Dniprop Reg Council SI DMA of MOH of Ukr Ch of Endocrinology, Dnipro
  - Medical Center of Limited Liability Company Medical Center Clinic of Family Medicine, Dnipro
  - Regional CH Dept of Endocrinology SHEI Ivano-Frankivsk NMU, Ivano-Frankivsk
  - CI Ivano-Frankivsk Reg Cl Card Center Dept of Chronic Ischemic Heart Dis SHEI Ivano-Frank NMU, Ivano-Frankivsk
  - Ivano-Frankivsk CCH Dept of Therapy #1 SHEI Ivano-Frankivsk NMU, Ivano-Frankivsk
  - CHI Kharkiv City Student Hosp Therap dept Nat Pharm Univer, Kharkiv
  - CNE Prof. O.O. Shalimov Kharkiv City Clinical Hospital #2 KCC, Kharkiv
  - GI L.T.Malaya Therapy National Institute of the NAMS of Ukraine, Kharkiv
  - State Institution LT Malaya Inst. of Ther. of AMS of Ukraine, Kharkiv
  - Railway Transport Kharkiv CH #1 of Healthcare Center Branch of PJSC Ukr Railway, Kharkiv
  - Railway Transport Kharkiv CH#1 of Healthcare Center Branch of PJSC Ukrainian Railway, Kharkiv
  - MC Doctor Alex Dept of General Practice-Family Medicine Kharkiv MA of PGE, Kharkiv
  - CNE City Clin Hosp #8 of KCC Dept of Therapy Kharkiv MA of PGE of MOHU, Kharkiv
  - CI Ye.Ye.Karabelesh Kherson City Clinical Hosp., Kherson
  - KCCC of Endocr Dept of General Endocrine Pathology O. O. Bogomolets NMU, Kyiv
  - Kyiv CCH #12 Dept of Therapy O.O.Bogomolets NMU, Kyiv
  - LLC Treatment and Diagnostic Center Adonis Plus, Kyiv
  - MC of PHEI Institute of General Practice - Family Medicine, Kyiv
  - Medical Center Blagomed Plus LLC, Kyiv
  - Med Center 'Ok!Clinic+' of International Institute of Clinical Trials LLC, Kyiv
  - MC of Subsidiary Production Unit Med Scient Pract Union Medbud of PJSc Holding Company Kyivmiskbud, Kyiv
  - Kyiv CH on Railway Transport #2 of Branch Center of Healthcare Public Company Ukr Railway, Kyiv
  - Med Center of Eurolab LLC Policlinic Outpatient Dept O.O.Bogomolets NMU, Kyiv
  - SI National Scientific Centre of Radiation Medicine of NAMSU, Kyiv
  - SI NSC M.D. Strazhesko Institute of Cardiology of NAMSU, Kyiv
  - SI NSС M.D. Strazhesko Institute of Cardiology of NAMSU, Kyiv
  - Department of Medical Services and Rehabilitation of State Joint Stock Holding Company Artem, Kyiv
  - Medical Center of Limited Liability Company Medical Center Concilium Medical, Kyiv
  - CI of Kyiv RC Regional Clinical Hospital #2, Kyiv
  - SI V.P.Komisarenko Institute of E&M of NAMSU, Kyiv
  - SI V.P.Komisarenko Institute of Endocrinology and Metabolism of NAMSU, Kyiv
  - Lviv Reg St Clin Treatment - Diagnostic Endocrin Center, Dept of Polyclinic, D.Galytskyy Lviv NMU, Lviv
  - Lviv Communal 4th City Clinical Hospital, Lviv
  - Center of Reconstructive & Restorative Medicine (University Clinic) of Odessa National Medical Uni, Odesa
  - CI Sumy City Clinical Hospital #1 Dept of Therapy Sumy SU Med Inst, Sumy
  - Ternopil City Municipal Hospital #2 Dept of Gastroenterology Ternopil I.Ya. Gorbachevskyi SMU, Ternopil
  - Transcarpathian Regional Clinical Cardiology Dispansery, Uzhhorod
  - Private Small Enterprise Medical Center Pulse, Vinnytsia
  - Vinnytsia RC Highly Special.Endocr.Center Dept of Therapy #2 M.I. Pyrogov NMU, Vinnytsia
  - National Pirogov Memorial Medical University, Vinnytsia
  - SRI of Invalid Rehabilitation (EST Complex) of Vinnytsia M.I.Pyrogov NMU MOHU, Vinnytsia
  - CI Zapor CCH#10 SI ZMA PGE Ch of therapy clin pharmacol & endocrin, Zaporizhzhia
  - CI Central City Hospital #1 of Zhytomyr, Zhytomyr
  - Zhytomyr regional clinical hospital n.a. O.F. Gerbachevskyy, Zhytomyr
- United Kingdom (21):
  - Synexus Thames, Reading, Berkshire
  - Mounts Bay Medical Ltd, Hayle, Cornwall
  - Oak Tree Surgery, Liskeard, Cornwall
  - The Alverton Practice, Penzance, Cornwall
  - Rame Medical Limited, Torpoint, Cornwall
  - Knowle House Surgery, Plymouth, Devon
  - Torbay Hospital, Torquay, Devon
  - Synexus Clinical Research North Tees, Stockton-on-Tees, Durham
  - Broomfield Hospital, Chelmsford, Essex
  - Barts Hospital, London, Greater London
  - Manchester Royal Infirmary, Manchester, Greater Manchester
  - Synexus Manchester Clinical Research Centre, Manchester, Greater Manchester
  - Waterloo Medical Centre, Blackpool, Lancashire
  - Synexus Lancashire Clinical Research Centre, Chorley, Lancashire
  - Synexus Merseyside Clinical Research Centre, Liverpool, Merseyside
  - Synexus Hexham General Hospital, Hexham, Northumberland
  - Synexus Wales Clinical Research Centre, Cardiff, South Glamorgan
  - Synexus Scotland Clinical Research Centre, Glasgow, Strathclyde
  - Ninewells Hospital, Dundee, Tayside Region
  - Synexus Birmingham Clinical Research Centre, Birmingham, West Midlands
  - Morriston Hospital, Swansea

REFERENCES:
- [Derived] Das Pradhan A, Glynn RJ, Fruchart JC, MacFadyen JG, Zaharris ES, Everett BM, Campbell SE, Oshima R, Amarenco P, Blom DJ, Brinton EA, Eckel RH, Elam MB, Felicio JS, Ginsberg HN, Goudev A, Ishibashi S, Joseph J, Kodama T, Koenig W, Leiter LA, Lorenzatti AJ, Mankovsky B, Marx N, Nordestgaard BG, Pall D, Ray KK, Santos RD, Soran H, Susekov A, Tendera M, Yokote K, Paynter NP, Buring JE, Libby P, Ridker PM; PROMINENT Investigators. Triglyceride Lowering with Pemafibrate to Reduce Cardiovascular Risk. N Engl J Med. 2022 Nov 24;387(21):1923-1934. doi: 10.1056/NEJMoa2210645. Epub 2022 Nov 5. PMID 36342113
- [Derived] Pradhan AD, Paynter NP, Everett BM, Glynn RJ, Amarenco P, Elam M, Ginsberg H, Hiatt WR, Ishibashi S, Koenig W, Nordestgaard BG, Fruchart JC, Libby P, Ridker PM. Rationale and design of the Pemafibrate to Reduce Cardiovascular Outcomes by Reducing Triglycerides in Patients with Diabetes (PROMINENT) study. Am Heart J. 2018 Dec;206:80-93. doi: 10.1016/j.ahj.2018.09.011. Epub 2018 Sep 29. PMID 30342298

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Prior to treatment, participants attended a Prescreening Visit, a Screening/Enrollment Visit and a Placebo Run-In Period. Eligible subjects who were compliant with study treatment during the Placebo Run-In Period returned for the Randomization Visit, at which time they were randomly allocated to receive either pemafibrate or a matching placebo tablet.
Groups:
- Pemafibrate: Participants receiving K-877 tablets administered twice daily.
- Placebo: Participants receiving Placebo matching tablet twice daily.
Period: Overall Study
Arm/Group | Pemafibrate | Placebo
Started | 5269 | 5275
Completed | 4647 | 4674
Not Completed | 622 | 601

BASELINE CHARACTERISTICS:
Population: The Intent to treat (ITT) population included all randomized subjects who received at least 1 dose of study treatment without GCP deviations.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pemafibrate | Placebo | Total
Number analyzed (Participants) | 5240 | 5257 | 10497
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.28 (8.524) | 63.56 (8.411) | 63.42 (8.468)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1443 | 1448 | 2891
  Male | 3797 | 3809 | 7606
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1014 | 1007 | 2021
  Not Hispanic or Latino | 4187 | 4213 | 8400
  Unknown or Not Reported | 39 | 37 | 76
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 4484 | 4549 | 9033
  Black or African American | 134 | 136 | 270
  American Indian or Alaska Native | 73 | 76 | 149
  Asian Indian | 97 | 80 | 177
  Bangladeshi | 0 | 3 | 3
  Chinese | 3 | 1 | 4
  Filipino | 2 | 5 | 7
  Japanese | 162 | 146 | 308
  Korean | 0 | 0 | 0
  Pakistani | 13 | 6 | 19
  Vietnamese | 1 | 0 | 1
  Other Asian | 13 | 10 | 23
  Native Hawaiian | 0 | 0 | 0
  Guamanian or Chamorro | 0 | 0 | 0
  Samoan | 0 | 0 | 0
  Other Pacific Islander | 1 | 0 | 1
  Multiracial | 29 | 32 | 61
  Other | 208 | 201 | 409
  Declined | 20 | 12 | 32
Cardiovascular Diseases and Risk Factors at Baseline [Count of Participants; unit: Participants] — To qualify for this study, subjects had to have type 2 diabetes (T2D) and a high risk for future cardiovascular (CV) events.
  Participants
    Statin Status: No | 220 | 219 | 439
    Statin Status: Yes | 5020 | 5038 | 10058
    Established CV Disease: No | 1695 | 1713 | 3408
    Established CV Disease: Yes | 3545 | 3544 | 7089

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With First Occurrence of 4-component Composite Primary Endpoint (Nonfatal MI, Nonfatal Ischemic Stroke, Coronary Revascularization, or CV Death)
Description: Number of participants experiencing their first occurrence of any component of the 4-component composite primary endpoint, which includes nonfatal myocardial infarction (MI), nonfatal ischemic stroke, coronary revascularization, or cardiovascular (CV) death. Each participant is counted only once, regardless of any subsequent events.
Time Frame: From Baseline to a Median of 3.3 Years
Population: Intention to treat population (ITT)
Measure: Number; unit: participants
Arm/Group | Pemafibrate | Placebo
Number analyzed (Participants) | 5240 | 5257
participants | 590 | 570
Statistical Analysis 1: Comparison: Pemafibrate vs Placebo; Test type: Superiority; Hazard Ratio (HR) = 1.03, 95% CI 2-sided [0.92 to 1.16]

2. Secondary Outcome: Number of Participants With First Occurrence of the 4-component Composite Secondary Endpoint (Nonfatal MI, Nonfatal Ischemic Stroke, Hospitalization for Unstable Angina Requiring Unplanned Coronary Revascularization, or CV Death)
Description: The 4-component composite secondary endpoints events are nonfatal myocardial infarction, nonfatal ischemic stroke, hospitalization for unstable angina requiring unplanned coronary revascularization, or cardiovascular death
Time Frame: From Baseline to a Median of 3.3 Years
Population: ITT population
Measure: Number; unit: participants
Arm/Group | Pemafibrate | Placebo
Number analyzed (Participants) | 5240 | 5257
participants | 447 | 427
Statistical Analysis 1: Comparison: Pemafibrate vs Placebo; Test type: Superiority; Hazard Ratio (HR) = 1.05, 95% CI 2-sided [0.92 to 1.20]

3. Secondary Outcome: Number of Participants With First Occurrence of the 3-component Composite Endpoint (Nonfatal Myocardial Infarction, Nonfatal Ischemic Stroke, or Cardiovascular Death)
Description: Number of Participants with First Occurrence of Composite Cardiovascular Events (nonfatal myocardial infarction, nonfatal ischemic stroke, or cardiovascular death)
Time Frame: From Baseline to a Median of 3.3 Years
Population: ITT population
Measure: Number; unit: participants
Arm/Group | Pemafibrate | Placebo
Number analyzed (Participants) | 5240 | 5257
participants | 396 | 386
Statistical Analysis 1: Comparison: Pemafibrate vs Placebo; Test type: Superiority; Hazard Ratio (HR) = 1.03, 95% CI 2-sided [0.89 to 1.18]

4. Secondary Outcome: Number of Participants With First Occurrence of Any Component of the Primary Endpoint or Hospitalization for Heart Failure
Description: Event is the first occurrence of any component of the composite endpoint of nonfatal myocardial infarction, nonfatal ischemic stroke, coronary revascularization, cardiovascular death, or hospitalization for heart failure
Time Frame: From Baseline to a Median of 3.3 Years
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Pemafibrate | Placebo
Number analyzed (Participants) | 5240 | 5257
participants | 670 | 645
Statistical Analysis 1: Comparison: Pemafibrate vs Placebo; Test type: Superiority; Hazard Ratio (HR) = 1.04, 95% CI 2-sided [0.93 to 1.16]

5. Secondary Outcome: Number of Participants With Occurrence of Any Component of the Primary Endpoint or All-Cause Mortality
Description: Event is the first occurrence of any component of the composite endpoint of nonfatal myocardial infarction, nonfatal ischemic stroke, coronary revascularization, cardiovascular death, or all-cause mortality.
Time Frame: From Baseline to a Median of 3.3 Years
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Pemafibrate | Placebo
Number analyzed (Participants) | 5240 | 5257
participants | 830 | 806
Statistical Analysis 1: Comparison: Pemafibrate vs Placebo; Test type: Superiority; Hazard Ratio (HR) = 1.03, 95% CI 2-sided [0.93 to 1.13]

6. Secondary Outcome: Total Number of Events of the 4-component Composite Primary Endpoint
Description: Total number of events for the 4-component composite primary endpoint, counting all occurrences, including multiple events in the same participant. The endpoint events include nonfatal myocardial infarction (MI), nonfatal ischemic stroke, coronary revascularization, and cardiovascular (CV) death.
Time Frame: From Baseline to a Median of 3.3 Years
Population: ITT Population
Measure: Number; unit: Events
Arm/Group | Pemafibrate | Placebo
Number analyzed (Participants) | 5240 | 5257
Events | 895 | 892
Statistical Analysis 1: Comparison: Pemafibrate vs Placebo; Test type: Superiority; Event Rate Ration = 0.99, 95% CI 2-sided [0.87 to 1.13]

7. Secondary Outcome: Number of Participants With First Occurrence of Any New or Worsening Peripheral Artery Disease (PAD)
Description: Any new or worsening Peripheral artery disease (PAD), defined as incidence of lower extremity revascularization, intermittent claudication, rest pain, lower extremity ischemic ulceration, or major amputation with either ankle-brachial index ≤ 0.9 or other diagnostic testing (eg, toe-brachial index, angiogram, or other imaging study)
Time Frame: From Baseline to a Median of 3.3 Years
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Pemafibrate | Placebo
Number analyzed (Participants) | 5240 | 5257
participants | 138 | 159
Statistical Analysis 1: Comparison: Pemafibrate vs Placebo; Test type: Superiority; Hazard Ratio (HR) = 0.87, 95% CI 2-sided [0.69 to 1.09]

8. Secondary Outcome: Number of Participants With First Occurrence of Nonfatal Myocardial Infarction
Time Frame: From Baseline to a Median of 3.3 Years
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Pemafibrate | Placebo
Number analyzed (Participants) | 5240 | 5257
participants | 210 | 182
Statistical Analysis 1: Comparison: Pemafibrate vs Placebo; Test type: Superiority; Hazard Ratio (HR) = 1.16, 95% CI 2-sided [0.95 to 1.41]

9. Secondary Outcome: Number of Participants With First Occurrence of Nonfatal Ischemic Stroke
Time Frame: From Baseline to a Median of 3.3 Years
Population: ITT population
Measure: Number; unit: participants
Arm/Group | Pemafibrate | Placebo
Number analyzed (Participants) | 5240 | 5257
participants | 96 | 106
Statistical Analysis 1: Comparison: Pemafibrate vs Placebo; Test type: Superiority; Hazard Ratio (HR) = 0.90, 95% CI 2-sided [0.69 to 1.19]

10. Secondary Outcome: Number of Participants With First Occurrence of Coronary Revascularization
Time Frame: From Baseline to a Median of 3.3 Years
Population: ITT population
Measure: Number; unit: participants
Arm/Group | Pemafibrate | Placebo
Number analyzed (Participants) | 5240 | 5257
participants | 340 | 347
Statistical Analysis 1: Comparison: Pemafibrate vs Placebo; Test type: Superiority; Hazard Ratio (HR) = 0.98, 95% CI 2-sided [0.84 to 1.14]

11. Secondary Outcome: Number of Participants With First Occurrence of Cardiovascular Death
Time Frame: From Baseline to a Median of 3.3 Years
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Pemafibrate | Placebo
Number analyzed (Participants) | 5240 | 5257
participants | 145 | 139
Statistical Analysis 1: Comparison: Pemafibrate vs Placebo; Test type: Superiority; Hazard Ratio (HR) = 1.04, 95% CI 2-sided [0.83 to 1.32]

12. Secondary Outcome: Number of Participants With First Occurrence of the 4-component Composite Endpoint by PPAR-α Gene Variant Subgroup (TT, CT, CC)
Description: Number of participants experiencing their first occurrence of any component of the 4-component composite primary endpoint (nonfatal myocardial infarction, nonfatal ischemic stroke, coronary revascularization, or cardiovascular death), reported as a subgroup analysis by PPAR-α gene variants (TT, CT, CC).
Time Frame: From Baseline to a Median of 3.3 Years
Population: This analysis includes participants from the intent-to-treat population who consented to genetic testing for the PPAR-α gene. Participants who did not provide consent for genetic testing are excluded from the numbers reported for this outcome measure.
Measure: Number; unit: Count of Participants
Arm/Group | Pemafibrate | Placebo
Number analyzed (Participants) | 2800 | 2841
Count of Participants
  TT variant: number analyzed (Participants) | 1011 | 973
  TT variant | 114 | 117
  CT variant: number analyzed (Participants) | 1312 | 1372
  CT variant | 177 | 156
  CC variant: number analyzed (Participants) | 477 | 496
  CC variant | 63 | 65
Statistical Analysis 1: Comparison: Pemafibrate vs Placebo; TT Variant; Test type: Superiority; Hazard Ratio (HR) = 0.97, 95% CI 2-sided [0.75 to 1.26]
Statistical Analysis 2: Comparison: Pemafibrate vs Placebo; CT Variant; Test type: Superiority; Hazard Ratio (HR) = 1.19, 95% CI 2-sided [0.96 to 1.47]
Statistical Analysis 3: Comparison: Pemafibrate vs Placebo; CC Variant; Test type: Superiority; Hazard Ratio (HR) = 0.98, 95% CI 2-sided [0.69 to 1.39]

13. Secondary Outcome: Percent Change From Baseline to Month 4 for Total Cholesterol (TC)
Time Frame: Baseline to Month 4
Population: * ITT population
  * The number of participants analyzed for the outcome measure may differ from the overall number of participants in each group. This discrepancy can be attributed to several factors, including:
    * Missing data: Some participants may have incomplete data due to factors such as missed visits, early withdrawal, refusal or inability to draw blood, or loss to follow-up.
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Pemafibrate | Placebo
Number analyzed (Participants) | 4859 | 4899
Percent Change | 5.235 (23.7683) | 4.562 (23.9991)
Statistical Analysis 1: Comparison: Pemafibrate vs Placebo; Test type: Superiority; p = 0.13496, ANCOVA

14. Secondary Outcome: Percent Change From Baseline to Month 4 for Fasting Triglycerides
Time Frame: Baseline to 4 Months
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Pemafibrate | Placebo
Number analyzed (Participants) | 4814 | 4848
Percent Change | -23.860 (49.2289) | 2.593 (60.6399)
Statistical Analysis 1: Comparison: Pemafibrate vs Placebo; Test type: Superiority; p < 0.001, ANCOVA

15. Secondary Outcome: Percent Change From Baseline to Month 4 for HDL - Cholesterol (HDL-C)
Time Frame: Baseline to Month 4
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Pemafibrate | Placebo
Number analyzed (Participants) | 4858 | 4896
Percent Change | 10.856 (24.7407) | 6.004 (21.7838)
Statistical Analysis 1: Comparison: Pemafibrate vs Placebo; Test type: Superiority; p < 0.001, ANCOVA

16. Secondary Outcome: Percent Change From Baseline to Month 4 for Calculated Non-HDL Cholesterol (Non-HDL-C)
Time Frame: Baseline to Month 4
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Pemafibrate | Placebo
Number analyzed (Participants) | 4858 | 4896
Percent Change | 5.219 (31.9262) | 5.502 (31.9739)
Statistical Analysis 1: Comparison: Pemafibrate vs Placebo; Test type: Superiority; p = 0.96689, ANCOVA

17. Secondary Outcome: Percent Change From Baseline to Month 4 for Calculated VLDL Cholesterol
Time Frame: Baseline to Month 4
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Pemafibrate | Placebo
Number analyzed (Participants) | 3841 | 3614
Percent Change | -22.788 (32.5741) | -1.601 (36.4352)
Statistical Analysis 1: Comparison: Pemafibrate vs Placebo; Test type: Superiority; p < 0.001, ANCOVA

18. Secondary Outcome: Percent Change From Baseline to Month 4 for Apolipoprotein A1 (ApoA1)
Time Frame: Baseline to Month 4
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Pemafibrate | Placebo
Number analyzed (Participants) | 4807 | 4847
Percent Change | 4.878 (19.3749) | 3.956 (18.5293)
Statistical Analysis 1: Comparison: Pemafibrate vs Placebo; Test type: Superiority; p = 0.09178, ANCOVA

19. Secondary Outcome: Percent Change From Baseline to Month 4 for Apolipoprotein CIII (ApoC3)
Time Frame: Baseline to Month 4
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Pemafibrate | Placebo
Number analyzed (Participants) | 4783 | 4808
Percent Change | -23.397 (31.5756) | 4.861 (56.0921)
Statistical Analysis 1: Comparison: Pemafibrate vs Placebo; Test type: Superiority; p < 0.001, ANCOVA

20. Secondary Outcome: Percent Change From Baseline to Month 4 for Apolipoprotein E (ApoE)
Time Frame: Baseline to Month 4
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Pemafibrate | Placebo
Number analyzed (Participants) | 4801 | 4842
Percent Change | -6.5201 (30.89475) | -0.5209 (31.79989)
Statistical Analysis 1: Comparison: Pemafibrate vs Placebo; Test type: Superiority; p < 0.001, ANCOVA

21. Secondary Outcome: Percent Change From Baseline to Month 6 for Non-fasting Remnant Cholesterol
Time Frame: Baseline to Month 6
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Pemafibrate | Placebo
Number analyzed (Participants) | 4614 | 4643
Percent Change | -21.27 (46.506) | 10.60 (54.029)
Statistical Analysis 1: Comparison: Pemafibrate vs Placebo; Test type: Superiority; p < 0.001, ANCOVA

ADVERSE EVENTS:
Time Frame: From Baseline to a Median of 3.3 Years
Description: Treatment emergent adverse events (TEAE) were any adverse event that occurred or worsened after the first dose of study treatment.
Arm/Group | Pemafibrate | Placebo
All-Cause Mortality (participants affected / at risk) | 308/5264 | 310/5274
Serious Adverse Events (participants affected / at risk) | 1715/5264 | 1663/5274
Other Adverse Events (participants affected / at risk) | 2817/5264 | 2883/5274
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pemafibrate (N=5264) | Placebo (N=5274)
Anaemia (Blood and lymphatic system disorders) | 10 | 10
Iron deficiency anaemia (Blood and lymphatic system disorders) | 5 | 6
Blood loss anaemia (Blood and lymphatic system disorders) | 3 | 3
Leukocytosis (Blood and lymphatic system disorders) | 0 | 3
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 2 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1
Hypochromic anaemia (Blood and lymphatic system disorders) | 2 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 2
Pancytopenia (Blood and lymphatic system disorders) | 2 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1
Anaemia of chronic disease (Blood and lymphatic system disorders) | 0 | 1
Hypercoagulation (Blood and lymphatic system disorders) | 0 | 1
Immune thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Microcytic anaemia (Blood and lymphatic system disorders) | 0 | 1
Normocytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Pernicious anaemia (Blood and lymphatic system disorders) | 0 | 1
Angina unstable (Cardiac disorders) | 97 | 95
Acute myocardial infarction (Cardiac disorders) | 97 | 93
Cardiac failure (Cardiac disorders) | 84 | 68
Angina pectoris (Cardiac disorders) | 69 | 59
Atrial fibrillation (Cardiac disorders) | 53 | 73
Coronary artery disease (Cardiac disorders) | 66 | 59
Myocardial infarction (Cardiac disorders) | 56 | 58
Cardiac failure congestive (Cardiac disorders) | 45 | 55
Coronary artery stenosis (Cardiac disorders) | 32 | 33
Cardiac failure acute (Cardiac disorders) | 19 | 16
Myocardial ischaemia (Cardiac disorders) | 13 | 22
Atrial flutter (Cardiac disorders) | 11 | 18
Cardiac failure chronic (Cardiac disorders) | 14 | 15
Ventricular tachycardia (Cardiac disorders) | 12 | 9
Arteriosclerosis coronary artery (Cardiac disorders) | 7 | 11
Coronary artery occlusion (Cardiac disorders) | 6 | 12
Acute left ventricular failure (Cardiac disorders) | 6 | 8
Acute coronary syndrome (Cardiac disorders) | 6 | 7
Atrioventricular block complete (Cardiac disorders) | 9 | 3
Aortic valve stenosis (Cardiac disorders) | 5 | 6
Bradycardia (Cardiac disorders) | 6 | 5
Left ventricular failure (Cardiac disorders) | 5 | 6
Arrhythmia (Cardiac disorders) | 7 | 3
Atrioventricular block second degree (Cardiac disorders) | 6 | 4
Cardiac arrest (Cardiac disorders) | 5 | 4
Sinus node dysfunction (Cardiac disorders) | 4 | 5
Supraventricular tachycardia (Cardiac disorders) | 7 | 1
Pericarditis (Cardiac disorders) | 3 | 3
Ventricular fibrillation (Cardiac disorders) | 4 | 2
Atrioventricular block (Cardiac disorders) | 1 | 4
Left ventricular dysfunction (Cardiac disorders) | 2 | 2
Palpitations (Cardiac disorders) | 1 | 3
Atrial tachycardia (Cardiac disorders) | 0 | 3
Bundle branch block left (Cardiac disorders) | 3 | 0
Cardio-respiratory arrest (Cardiac disorders) | 3 | 0
Ischaemic cardiomyopathy (Cardiac disorders) | 3 | 0
Ventricular extrasystoles (Cardiac disorders) | 1 | 2
Aortic valve incompetence (Cardiac disorders) | 0 | 2
Atrial thrombosis (Cardiac disorders) | 1 | 1
Cardiac ventricular thrombosis (Cardiac disorders) | 1 | 1
Coronary artery insufficiency (Cardiac disorders) | 1 | 1
Mitral valve stenosis (Cardiac disorders) | 1 | 1
Myocarditis (Cardiac disorders) | 1 | 1
Right ventricular failure (Cardiac disorders) | 0 | 2
Sinus arrest (Cardiac disorders) | 1 | 1
Sinus bradycardia (Cardiac disorders) | 2 | 0
Supraventricular extrasystoles (Cardiac disorders) | 2 | 0
Aortic valve calcification (Cardiac disorders) | 1 | 0
Aortic valve disease (Cardiac disorders) | 1 | 0
Arteriospasm coronary (Cardiac disorders) | 1 | 0
Atrioventricular block first degree (Cardiac disorders) | 1 | 0
Cardiac aneurysm (Cardiac disorders) | 0 | 1
Cardiac tamponade (Cardiac disorders) | 0 | 1
Cardiogenic shock (Cardiac disorders) | 0 | 1
Cardiomyopathy (Cardiac disorders) | 1 | 0
Cardiorenal syndrome (Cardiac disorders) | 0 | 1
Cardiovascular disorder (Cardiac disorders) | 0 | 1
Chronic coronary syndrome (Cardiac disorders) | 0 | 1
Conduction disorder (Cardiac disorders) | 1 | 0
Congestive cardiomyopathy (Cardiac disorders) | 1 | 0
Cor pulmonale acute (Cardiac disorders) | 0 | 1
Coronary artery dissection (Cardiac disorders) | 1 | 0
Coronary artery perforation (Cardiac disorders) | 1 | 0
Coronary artery thrombosis (Cardiac disorders) | 0 | 1
Degenerative aortic valve disease (Cardiac disorders) | 1 | 0
Hypertensive heart disease (Cardiac disorders) | 0 | 1
Low cardiac output syndrome (Cardiac disorders) | 1 | 0
Microvascular coronary artery disease (Cardiac disorders) | 0 | 1
Mitral valve incompetence (Cardiac disorders) | 1 | 0
Nodal rhythm (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0
Postinfarction angina (Cardiac disorders) | 0 | 1
Prinzmetal angina (Cardiac disorders) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 1 | 0
Stress cardiomyopathy (Cardiac disorders) | 0 | 1
Tachyarrhythmia (Cardiac disorders) | 1 | 0
Ventricular arrhythmia (Cardiac disorders) | 1 | 0
Hypertrophic cardiomyopathy (Congenital, familial and genetic disorders) | 1 | 1
Rathke's cleft cyst (Congenital, familial and genetic disorders) | 1 | 1
Congenital megaureter (Congenital, familial and genetic disorders) | 0 | 1
Gastrointestinal arteriovenous malformation (Congenital, familial and genetic disorders) | 0 | 1
Hydrocele (Congenital, familial and genetic disorders) | 0 | 1
Keratosis follicular (Congenital, familial and genetic disorders) | 0 | 1
Oesophageal cyst (Congenital, familial and genetic disorders) | 1 | 0
Skeletal dysplasia (Congenital, familial and genetic disorders) | 0 | 1
Venous angioma of brain (Congenital, familial and genetic disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 4 | 2
Acute vestibular syndrome (Ear and labyrinth disorders) | 0 | 1
Sudden hearing loss (Ear and labyrinth disorders) | 1 | 0
Vestibular disorder (Ear and labyrinth disorders) | 0 | 1
Goitre (Endocrine disorders) | 2 | 2
Primary hyperaldosteronism (Endocrine disorders) | 2 | 0
Hyperparathyroidism (Endocrine disorders) | 0 | 1
Hyperparathyroidism primary (Endocrine disorders) | 1 | 0
Hyperthyroidism (Endocrine disorders) | 1 | 0
Thyroid mass (Endocrine disorders) | 0 | 1
Cataract (Eye disorders) | 15 | 13
Retinal detachment (Eye disorders) | 5 | 1
Vitreous haemorrhage (Eye disorders) | 3 | 1
Glaucoma (Eye disorders) | 3 | 0
Strabismus (Eye disorders) | 1 | 1
Tractional retinal detachment (Eye disorders) | 2 | 0
Cataract nuclear (Eye disorders) | 1 | 0
Diabetic retinopathy (Eye disorders) | 1 | 0
Diplopia (Eye disorders) | 0 | 1
Dry eye (Eye disorders) | 1 | 0
Exophthalmos (Eye disorders) | 0 | 1
Iridocele (Eye disorders) | 1 | 0
Iris neovascularisation (Eye disorders) | 1 | 0
Macular fibrosis (Eye disorders) | 1 | 0
Macular hole (Eye disorders) | 1 | 0
Papilloedema (Eye disorders) | 0 | 1
Retinal tear (Eye disorders) | 1 | 0
Uveitis (Eye disorders) | 0 | 1
Visual acuity reduced (Eye disorders) | 1 | 0
Vitreoretinal traction syndrome (Eye disorders) | 1 | 0
Vitreous detachment (Eye disorders) | 1 | 0
Vitreous disorder (Eye disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 15 | 12
Pancreatitis acute (Gastrointestinal disorders) | 16 | 10
Inguinal hernia (Gastrointestinal disorders) | 8 | 5
Abdominal pain (Gastrointestinal disorders) | 4 | 7
Small intestinal obstruction (Gastrointestinal disorders) | 4 | 6
Large intestine polyp (Gastrointestinal disorders) | 5 | 4
Gastritis (Gastrointestinal disorders) | 5 | 3
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 6
Diarrhoea (Gastrointestinal disorders) | 1 | 6
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 4 | 3
Pancreatitis (Gastrointestinal disorders) | 5 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 4 | 2
Intestinal obstruction (Gastrointestinal disorders) | 2 | 4
Gastritis erosive (Gastrointestinal disorders) | 1 | 4
Obstructive pancreatitis (Gastrointestinal disorders) | 2 | 3
Vomiting (Gastrointestinal disorders) | 3 | 2
Colitis (Gastrointestinal disorders) | 3 | 1
Constipation (Gastrointestinal disorders) | 3 | 1
Gastric ulcer (Gastrointestinal disorders) | 1 | 3
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 3
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 2 | 2
Oesophageal spasm (Gastrointestinal disorders) | 1 | 3
Pancreatitis chronic (Gastrointestinal disorders) | 1 | 3
Umbilical hernia (Gastrointestinal disorders) | 2 | 2
Anal fistula (Gastrointestinal disorders) | 2 | 1
Colitis ulcerative (Gastrointestinal disorders) | 2 | 1
Diverticulum (Gastrointestinal disorders) | 2 | 1
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 2 | 1
Duodenal ulcer (Gastrointestinal disorders) | 3 | 0
Duodenitis (Gastrointestinal disorders) | 2 | 1
Ileus (Gastrointestinal disorders) | 1 | 2
Incarcerated umbilical hernia (Gastrointestinal disorders) | 1 | 2
Intestinal ischaemia (Gastrointestinal disorders) | 3 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 2
Abdominal hernia (Gastrointestinal disorders) | 2 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0
Ascites (Gastrointestinal disorders) | 1 | 1
Colitis ischaemic (Gastrointestinal disorders) | 1 | 1
Crohn's disease (Gastrointestinal disorders) | 1 | 1
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 2 | 0
Diverticulum intestinal (Gastrointestinal disorders) | 1 | 1
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 1
Dysphagia (Gastrointestinal disorders) | 2 | 0
Enterocolitis (Gastrointestinal disorders) | 2 | 0
Faecaloma (Gastrointestinal disorders) | 0 | 2
Gastrointestinal disorder (Gastrointestinal disorders) | 1 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 1
Hiatus hernia (Gastrointestinal disorders) | 2 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 1 | 1
Incarcerated inguinal hernia (Gastrointestinal disorders) | 1 | 1
Intestinal perforation (Gastrointestinal disorders) | 0 | 2
Mechanical ileus (Gastrointestinal disorders) | 1 | 1
Mesenteric artery stenosis (Gastrointestinal disorders) | 0 | 2
Oesophageal stenosis (Gastrointestinal disorders) | 2 | 0
Proctitis (Gastrointestinal disorders) | 1 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 1
Abdominal incarcerated hernia (Gastrointestinal disorders) | 0 | 1
Anal haemorrhage (Gastrointestinal disorders) | 1 | 0
Anal skin tags (Gastrointestinal disorders) | 0 | 1
Anal stenosis (Gastrointestinal disorders) | 0 | 1
Barrett's oesophagus (Gastrointestinal disorders) | 1 | 0
Chronic gastritis (Gastrointestinal disorders) | 0 | 1
Diverticular perforation (Gastrointestinal disorders) | 1 | 0
Duodenal perforation (Gastrointestinal disorders) | 0 | 1
Duodenal ulcer perforation (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Enteritis (Gastrointestinal disorders) | 0 | 1
Eosinophilic oesophagitis (Gastrointestinal disorders) | 1 | 0
Epigastric discomfort (Gastrointestinal disorders) | 0 | 1
Gastric disorder (Gastrointestinal disorders) | 0 | 1
Gastric ulcer perforation (Gastrointestinal disorders) | 1 | 0
Gastroduodenal haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrointestinal toxicity (Gastrointestinal disorders) | 0 | 1
Gastrointestinal vascular malformation haemorrhagic (Gastrointestinal disorders) | 1 | 0
Gastrointestinal wall thickening (Gastrointestinal disorders) | 0 | 1
Haematochezia (Gastrointestinal disorders) | 1 | 0
Inguinal hernia strangulated (Gastrointestinal disorders) | 1 | 0
Intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Intestinal mass (Gastrointestinal disorders) | 1 | 0
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 1
Large intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 0 | 1
Melaena (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Obstruction gastric (Gastrointestinal disorders) | 0 | 1
Oedematous pancreatitis (Gastrointestinal disorders) | 1 | 0
Oesophageal achalasia (Gastrointestinal disorders) | 1 | 0
Oesophageal obstruction (Gastrointestinal disorders) | 0 | 1
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0
Peptic ulcer (Gastrointestinal disorders) | 0 | 1
Pneumoretroperitoneum (Gastrointestinal disorders) | 0 | 1
Rectal polyp (Gastrointestinal disorders) | 1 | 0
Rectal prolapse (Gastrointestinal disorders) | 1 | 0
Retroperitoneal effusion (Gastrointestinal disorders) | 1 | 0
Salivary gland mass (Gastrointestinal disorders) | 0 | 1
Short-bowel syndrome (Gastrointestinal disorders) | 1 | 0
Small intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Small intestinal perforation (Gastrointestinal disorders) | 1 | 0
Small intestine ulcer (Gastrointestinal disorders) | 1 | 0
Splenic artery aneurysm (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0
Subileus (Gastrointestinal disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 30 | 38
Chest pain (General disorders) | 5 | 10
Vascular stent stenosis (General disorders) | 9 | 5
Asthenia (General disorders) | 6 | 2
Multiple organ dysfunction syndrome (General disorders) | 3 | 5
Pyrexia (General disorders) | 3 | 3
Oedema peripheral (General disorders) | 2 | 2
Fatigue (General disorders) | 0 | 3
Gait disturbance (General disorders) | 1 | 1
Impaired healing (General disorders) | 0 | 2
Pain (General disorders) | 1 | 1
Vascular device occlusion (General disorders) | 1 | 1
Catheter site inflammation (General disorders) | 0 | 1
Chest discomfort (General disorders) | 1 | 0
Drug intolerance (General disorders) | 1 | 0
Exercise tolerance decreased (General disorders) | 1 | 0
Hernia pain (General disorders) | 0 | 1
Localised oedema (General disorders) | 1 | 0
Malaise (General disorders) | 1 | 0
Peripheral swelling (General disorders) | 0 | 1
Physical deconditioning (General disorders) | 0 | 1
Prosthetic cardiac valve stenosis (General disorders) | 1 | 0
Stenosis (General disorders) | 1 | 0
Strangulated hernia (General disorders) | 1 | 0
Systemic inflammatory response syndrome (General disorders) | 1 | 0
Vascular stent thrombosis (General disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 23 | 14
Cholecystitis (Hepatobiliary disorders) | 15 | 15
Cholecystitis acute (Hepatobiliary disorders) | 15 | 8
Bile duct stone (Hepatobiliary disorders) | 4 | 2
Biliary obstruction (Hepatobiliary disorders) | 1 | 4
Cholecystitis chronic (Hepatobiliary disorders) | 2 | 2
Hepatic cirrhosis (Hepatobiliary disorders) | 3 | 1
Jaundice cholestatic (Hepatobiliary disorders) | 2 | 2
Biliary colic (Hepatobiliary disorders) | 1 | 1
Cholangitis (Hepatobiliary disorders) | 2 | 0
Hepatic mass (Hepatobiliary disorders) | 1 | 1
Nonalcoholic fatty liver disease (Hepatobiliary disorders) | 1 | 1
Acute hepatic failure (Hepatobiliary disorders) | 1 | 0
Cholangitis acute (Hepatobiliary disorders) | 0 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 0
Gallbladder oedema (Hepatobiliary disorders) | 1 | 0
Hepatic fibrosis (Hepatobiliary disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1
Hepatic steatosis (Hepatobiliary disorders) | 0 | 1
Hepatitis cholestatic (Hepatobiliary disorders) | 0 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Non-alcoholic steatohepatitis (Hepatobiliary disorders) | 1 | 0
Anaphylactic reaction (Immune system disorders) | 4 | 0
Amyloidosis (Immune system disorders) | 1 | 0
Contrast media allergy (Immune system disorders) | 0 | 1
Cytokine storm (Immune system disorders) | 0 | 1
Food allergy (Immune system disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 1
Sarcoidosis (Immune system disorders) | 0 | 1
COVID-19 pneumonia (Infections and infestations) | 95 | 91
Pneumonia (Infections and infestations) | 82 | 87
COVID-19 (Infections and infestations) | 57 | 50
Coronavirus infection (Infections and infestations) | 42 | 32
Cellulitis (Infections and infestations) | 30 | 28
Sepsis (Infections and infestations) | 31 | 25
Urinary tract infection (Infections and infestations) | 20 | 35
Osteomyelitis (Infections and infestations) | 16 | 17
Diverticulitis (Infections and infestations) | 14 | 8
Gastroenteritis (Infections and infestations) | 8 | 13
Appendicitis (Infections and infestations) | 10 | 10
Erysipelas (Infections and infestations) | 7 | 12
Urosepsis (Infections and infestations) | 7 | 12
Influenza (Infections and infestations) | 6 | 9
Gangrene (Infections and infestations) | 9 | 5
Pyelonephritis (Infections and infestations) | 6 | 7
Septic shock (Infections and infestations) | 7 | 5
Bronchitis (Infections and infestations) | 5 | 6
Lower respiratory tract infection (Infections and infestations) | 8 | 3
Escherichia sepsis (Infections and infestations) | 5 | 5
Localised infection (Infections and infestations) | 5 | 5
Cystitis (Infections and infestations) | 2 | 6
Device related infection (Infections and infestations) | 5 | 3
Diabetic foot infection (Infections and infestations) | 4 | 4
Pyelonephritis acute (Infections and infestations) | 2 | 6
Wound infection (Infections and infestations) | 4 | 4
Abscess limb (Infections and infestations) | 3 | 4
Bacteraemia (Infections and infestations) | 4 | 3
Anal abscess (Infections and infestations) | 4 | 2
Cholecystitis infective (Infections and infestations) | 3 | 3
Clostridium difficile colitis (Infections and infestations) | 4 | 2
Escherichia urinary tract infection (Infections and infestations) | 1 | 5
Post procedural infection (Infections and infestations) | 4 | 2
Herpes zoster (Infections and infestations) | 2 | 3
Pneumonia bacterial (Infections and infestations) | 1 | 4
Postoperative wound infection (Infections and infestations) | 2 | 3
Bacterial sepsis (Infections and infestations) | 2 | 2
Infection (Infections and infestations) | 4 | 0
Pneumonia viral (Infections and infestations) | 1 | 3
Pulmonary sepsis (Infections and infestations) | 4 | 0
Pyelonephritis chronic (Infections and infestations) | 2 | 2
Streptococcal sepsis (Infections and infestations) | 3 | 1
Abdominal abscess (Infections and infestations) | 2 | 1
Arthritis bacterial (Infections and infestations) | 1 | 2
Arthritis infective (Infections and infestations) | 1 | 2
Atypical pneumonia (Infections and infestations) | 1 | 2
Bacterial pyelonephritis (Infections and infestations) | 2 | 1
Breast abscess (Infections and infestations) | 0 | 3
Dengue fever (Infections and infestations) | 0 | 3
Diabetic gangrene (Infections and infestations) | 2 | 1
Empyema (Infections and infestations) | 1 | 2
Escherichia bacteraemia (Infections and infestations) | 2 | 1
Fournier's gangrene (Infections and infestations) | 0 | 3
Gastroenteritis bacterial (Infections and infestations) | 3 | 0
Helicobacter gastritis (Infections and infestations) | 3 | 0
Intervertebral discitis (Infections and infestations) | 1 | 2
Lung abscess (Infections and infestations) | 2 | 1
Pneumococcal sepsis (Infections and infestations) | 2 | 1
Subcutaneous abscess (Infections and infestations) | 0 | 3
Upper respiratory tract infection (Infections and infestations) | 0 | 3
Appendicitis perforated (Infections and infestations) | 2 | 0
Bursitis infective (Infections and infestations) | 2 | 0
Cellulitis staphylococcal (Infections and infestations) | 1 | 1
Cellulitis streptococcal (Infections and infestations) | 1 | 1
Clostridium difficile infection (Infections and infestations) | 1 | 1
Emphysematous cystitis (Infections and infestations) | 1 | 1
Escherichia infection (Infections and infestations) | 1 | 1
Gastroenteritis rotavirus (Infections and infestations) | 1 | 1
Gastroenteritis viral (Infections and infestations) | 1 | 1
Groin abscess (Infections and infestations) | 1 | 1
Implant site infection (Infections and infestations) | 2 | 0
Infected skin ulcer (Infections and infestations) | 1 | 1
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 | 1
Klebsiella sepsis (Infections and infestations) | 2 | 0
Liver abscess (Infections and infestations) | 2 | 0
Lyme disease (Infections and infestations) | 1 | 1
Mastoiditis (Infections and infestations) | 1 | 1
Mediastinitis (Infections and infestations) | 0 | 2
Otitis externa (Infections and infestations) | 0 | 2
Pelvic abscess (Infections and infestations) | 0 | 2
Peritonitis (Infections and infestations) | 1 | 1
Rectal abscess (Infections and infestations) | 1 | 1
Respiratory syncytial virus infection (Infections and infestations) | 2 | 0
Respiratory tract infection (Infections and infestations) | 2 | 0
Sinusitis (Infections and infestations) | 2 | 0
Soft tissue infection (Infections and infestations) | 0 | 2
Staphylococcal bacteraemia (Infections and infestations) | 1 | 1
Staphylococcal osteomyelitis (Infections and infestations) | 2 | 0
Staphylococcal sepsis (Infections and infestations) | 1 | 1
Urinary tract infection bacterial (Infections and infestations) | 1 | 1
Urinary tract infection pseudomonal (Infections and infestations) | 0 | 2
Wound sepsis (Infections and infestations) | 1 | 1
Abdominal sepsis (Infections and infestations) | 1 | 0
Abdominal wall abscess (Infections and infestations) | 1 | 0
Abscess neck (Infections and infestations) | 1 | 0
Actinomycotic pulmonary infection (Infections and infestations) | 0 | 1
Acute hepatitis B (Infections and infestations) | 0 | 1
Alpha haemolytic streptococcal infection (Infections and infestations) | 1 | 0
Anorectal cellulitis (Infections and infestations) | 1 | 0
Bacterial tracheitis (Infections and infestations) | 0 | 1
Bartholinitis (Infections and infestations) | 1 | 0
Brain abscess (Infections and infestations) | 1 | 0
Bronchitis viral (Infections and infestations) | 1 | 0
Bullous erysipelas (Infections and infestations) | 0 | 1
Candida infection (Infections and infestations) | 0 | 1
Chest wall abscess (Infections and infestations) | 0 | 1
Chikungunya virus infection (Infections and infestations) | 1 | 0
Cholangitis infective (Infections and infestations) | 1 | 0
Chronic sinusitis (Infections and infestations) | 0 | 1
Clostridium colitis (Infections and infestations) | 1 | 0
Cyclosporidium infection (Infections and infestations) | 1 | 0
Dengue haemorrhagic fever (Infections and infestations) | 1 | 0
Diverticulitis intestinal perforated (Infections and infestations) | 0 | 1
Ear infection (Infections and infestations) | 1 | 0
Ear infection viral (Infections and infestations) | 0 | 1
Eczema herpeticum (Infections and infestations) | 0 | 1
Eczema infected (Infections and infestations) | 1 | 0
Emphysematous pyelonephritis (Infections and infestations) | 1 | 0
Enterobacter pneumonia (Infections and infestations) | 0 | 1
Enterococcal bacteraemia (Infections and infestations) | 1 | 0
Enterococcal infection (Infections and infestations) | 0 | 1
Epididymitis (Infections and infestations) | 0 | 1
Epstein-Barr virus infection (Infections and infestations) | 1 | 0
Extradural abscess (Infections and infestations) | 0 | 1
Gallbladder empyema (Infections and infestations) | 1 | 0
Gastric infection (Infections and infestations) | 1 | 0
Graft infection (Infections and infestations) | 0 | 1
Groin infection (Infections and infestations) | 0 | 1
Haematoma infection (Infections and infestations) | 1 | 0
HCoV-HKU1 infection (Infections and infestations) | 1 | 0
Hepatitis B (Infections and infestations) | 1 | 0
Hepatitis viral (Infections and infestations) | 1 | 0
Herpes zoster oticus (Infections and infestations) | 1 | 0
Infected dermal cyst (Infections and infestations) | 1 | 0
Infectious mononucleosis (Infections and infestations) | 1 | 0
Infectious pleural effusion (Infections and infestations) | 0 | 1
Intestinal sepsis (Infections and infestations) | 1 | 0
Klebsiella infection (Infections and infestations) | 1 | 0
Labyrinthitis (Infections and infestations) | 1 | 0
Large intestine infection (Infections and infestations) | 1 | 0
Lymph node tuberculosis (Infections and infestations) | 0 | 1
Mastitis (Infections and infestations) | 1 | 0
Meningococcal infection (Infections and infestations) | 1 | 0
Meningoencephalitis bacterial (Infections and infestations) | 1 | 0
Metapneumovirus pneumonia (Infections and infestations) | 1 | 0
Myelitis (Infections and infestations) | 0 | 1
Necrotising fasciitis (Infections and infestations) | 0 | 1
Neutropenic sepsis (Infections and infestations) | 1 | 0
Oesophageal candidiasis (Infections and infestations) | 0 | 1
Ophthalmic herpes zoster (Infections and infestations) | 1 | 0
Oral candidiasis (Infections and infestations) | 0 | 1
Orchitis (Infections and infestations) | 0 | 1
Osteomyelitis bacterial (Infections and infestations) | 1 | 0
Otitis media acute (Infections and infestations) | 0 | 1
Otitis media chronic (Infections and infestations) | 0 | 1
Paronychia (Infections and infestations) | 1 | 0
Perichondritis (Infections and infestations) | 0 | 1
Periorbital cellulitis (Infections and infestations) | 1 | 0
Peritonsillar abscess (Infections and infestations) | 0 | 1
Pneumonia fungal (Infections and infestations) | 1 | 0
Pneumonia legionella (Infections and infestations) | 1 | 0
Pneumonia necrotising (Infections and infestations) | 0 | 1
Pneumonia pneumococcal (Infections and infestations) | 1 | 0
Pneumonia pseudomonal (Infections and infestations) | 0 | 1
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 | 1
Post procedural sepsis (Infections and infestations) | 0 | 1
Pseudomembranous colitis (Infections and infestations) | 1 | 0
Pseudomonas infection (Infections and infestations) | 1 | 0
Pulmonary tuberculosis (Infections and infestations) | 1 | 0
Respiratory tract infection bacterial (Infections and infestations) | 0 | 1
Rhinitis (Infections and infestations) | 0 | 1
Septic arthritis staphylococcal (Infections and infestations) | 0 | 1
Serratia infection (Infections and infestations) | 0 | 1
Sialoadenitis (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 1 | 0
Splenic abscess (Infections and infestations) | 1 | 0
Staphylococcal infection (Infections and infestations) | 0 | 1
Streptococcal abscess (Infections and infestations) | 0 | 1
Streptococcal bacteraemia (Infections and infestations) | 1 | 0
Streptococcal infection (Infections and infestations) | 0 | 1
Tooth abscess (Infections and infestations) | 1 | 0
Tooth infection (Infections and infestations) | 0 | 1
Tracheobronchitis (Infections and infestations) | 0 | 1
Urinary tract infection enterococcal (Infections and infestations) | 0 | 1
Vaginal infection (Infections and infestations) | 0 | 1
Vascular device infection (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 1 | 0
Viral sepsis (Infections and infestations) | 1 | 0
Wound infection staphylococcal (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 9 | 8
Ankle fracture (Injury, poisoning and procedural complications) | 8 | 6
Hip fracture (Injury, poisoning and procedural complications) | 7 | 6
Femur fracture (Injury, poisoning and procedural complications) | 5 | 6
Limb injury (Injury, poisoning and procedural complications) | 5 | 5
Lower limb fracture (Injury, poisoning and procedural complications) | 6 | 3
Rib fracture (Injury, poisoning and procedural complications) | 8 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 6 | 2
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 4 | 4
Subdural haematoma (Injury, poisoning and procedural complications) | 4 | 4
Tendon rupture (Injury, poisoning and procedural complications) | 3 | 5
Toxicity to various agents (Injury, poisoning and procedural complications) | 7 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 6 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 3 | 4
Concussion (Injury, poisoning and procedural complications) | 5 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 2 | 4
Hand fracture (Injury, poisoning and procedural complications) | 3 | 3
Head injury (Injury, poisoning and procedural complications) | 2 | 4
Coronary artery restenosis (Injury, poisoning and procedural complications) | 2 | 3
Craniocerebral injury (Injury, poisoning and procedural complications) | 2 | 3
Intentional overdose (Injury, poisoning and procedural complications) | 2 | 3
Meniscus injury (Injury, poisoning and procedural complications) | 1 | 4
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 3 | 2
Wrist fracture (Injury, poisoning and procedural complications) | 2 | 3
Contusion (Injury, poisoning and procedural complications) | 2 | 2
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 3
Overdose (Injury, poisoning and procedural complications) | 3 | 1
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 3
Procedural pain (Injury, poisoning and procedural complications) | 1 | 3
Radius fracture (Injury, poisoning and procedural complications) | 1 | 3
Tibia fracture (Injury, poisoning and procedural complications) | 2 | 2
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 2 | 2
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 2 | 1
Chest injury (Injury, poisoning and procedural complications) | 3 | 0
Incisional hernia (Injury, poisoning and procedural complications) | 1 | 2
Postoperative wound complication (Injury, poisoning and procedural complications) | 2 | 1
Skin laceration (Injury, poisoning and procedural complications) | 1 | 2
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 1
Animal bite (Injury, poisoning and procedural complications) | 2 | 0
Arterial injury (Injury, poisoning and procedural complications) | 2 | 0
Burns third degree (Injury, poisoning and procedural complications) | 2 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 2
Injury (Injury, poisoning and procedural complications) | 2 | 0
Jaw fracture (Injury, poisoning and procedural complications) | 2 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 2 | 0
Muscle rupture (Injury, poisoning and procedural complications) | 1 | 1
Post procedural myocardial infarction (Injury, poisoning and procedural complications) | 2 | 0
Scapula fracture (Injury, poisoning and procedural complications) | 2 | 0
Skull fracture (Injury, poisoning and procedural complications) | 0 | 2
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 | 1
Traumatic haematoma (Injury, poisoning and procedural complications) | 1 | 1
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 1 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 1
Accident at work (Injury, poisoning and procedural complications) | 0 | 1
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 | 1
Adjacent segment degeneration (Injury, poisoning and procedural complications) | 0 | 1
Arteriovenous fistula maturation failure (Injury, poisoning and procedural complications) | 1 | 0
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0
Bite (Injury, poisoning and procedural complications) | 0 | 1
Bone contusion (Injury, poisoning and procedural complications) | 0 | 1
Bone fissure (Injury, poisoning and procedural complications) | 1 | 0
Brain contusion (Injury, poisoning and procedural complications) | 0 | 1
Burns second degree (Injury, poisoning and procedural complications) | 1 | 0
Cardiac contusion (Injury, poisoning and procedural complications) | 1 | 0
Cardiac function disturbance postoperative (Injury, poisoning and procedural complications) | 1 | 0
Cartilage injury (Injury, poisoning and procedural complications) | 0 | 1
Cataract operation complication (Injury, poisoning and procedural complications) | 1 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 1 | 0
Costal cartilage fracture (Injury, poisoning and procedural complications) | 1 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 1
Fracture displacement (Injury, poisoning and procedural complications) | 0 | 1
Gun shot wound (Injury, poisoning and procedural complications) | 1 | 0
Heat exhaustion (Injury, poisoning and procedural complications) | 0 | 1
Heat illness (Injury, poisoning and procedural complications) | 0 | 1
Incision site impaired healing (Injury, poisoning and procedural complications) | 0 | 1
Intervertebral disc injury (Injury, poisoning and procedural complications) | 0 | 1
Joint injury (Injury, poisoning and procedural complications) | 1 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0
Lip injury (Injury, poisoning and procedural complications) | 1 | 0
Multiple fractures (Injury, poisoning and procedural complications) | 0 | 1
Multiple injuries (Injury, poisoning and procedural complications) | 0 | 1
Osteophyte fracture (Injury, poisoning and procedural complications) | 0 | 1
Patella fracture (Injury, poisoning and procedural complications) | 0 | 1
Peripheral artery restenosis (Injury, poisoning and procedural complications) | 0 | 1
Periprosthetic fracture (Injury, poisoning and procedural complications) | 1 | 0
Pneumothorax traumatic (Injury, poisoning and procedural complications) | 1 | 0
Post concussion syndrome (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Postoperative renal failure (Injury, poisoning and procedural complications) | 0 | 1
Postoperative respiratory failure (Injury, poisoning and procedural complications) | 1 | 0
Postoperative thoracic procedure complication (Injury, poisoning and procedural complications) | 1 | 0
Procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Procedural pneumothorax (Injury, poisoning and procedural complications) | 0 | 1
Seroma (Injury, poisoning and procedural complications) | 1 | 0
Shunt thrombosis (Injury, poisoning and procedural complications) | 1 | 0
Soft tissue injury (Injury, poisoning and procedural complications) | 1 | 0
Spinal column injury (Injury, poisoning and procedural complications) | 0 | 1
Spinal cord injury (Injury, poisoning and procedural complications) | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0
Stress fracture (Injury, poisoning and procedural complications) | 0 | 1
Tendon injury (Injury, poisoning and procedural complications) | 1 | 0
Traumatic fracture (Injury, poisoning and procedural complications) | 1 | 0
Traumatic haemothorax (Injury, poisoning and procedural complications) | 0 | 1
Ulna fracture (Injury, poisoning and procedural complications) | 0 | 1
Vascular pseudoaneurysm ruptured (Injury, poisoning and procedural complications) | 1 | 0
VIth nerve injury (Injury, poisoning and procedural complications) | 1 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 0
Wound complication (Injury, poisoning and procedural complications) | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 1
Wound necrosis (Injury, poisoning and procedural complications) | 0 | 1
SARS-CoV-2 test positive (Investigations) | 1 | 8
Blood glucose increased (Investigations) | 4 | 2
Blood pressure increased (Investigations) | 3 | 1
Catheterisation cardiac (Investigations) | 2 | 1
Alanine aminotransferase increased (Investigations) | 1 | 1
Blood urea increased (Investigations) | 1 | 1
Ejection fraction decreased (Investigations) | 2 | 0
Glomerular filtration rate decreased (Investigations) | 0 | 2
Liver function test increased (Investigations) | 0 | 2
Prostatic specific antigen increased (Investigations) | 0 | 2
Transaminases increased (Investigations) | 1 | 1
Albumin urine present (Investigations) | 0 | 1
Anticoagulation drug level above therapeutic (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 0 | 1
Blood iron decreased (Investigations) | 1 | 0
Cardioactive drug level below therapeutic (Investigations) | 0 | 1
Device function test (Investigations) | 1 | 0
Electrocardiogram ST segment elevation (Investigations) | 1 | 0
Glycosylated haemoglobin increased (Investigations) | 0 | 1
Heart rate increased (Investigations) | 1 | 0
Heart rate irregular (Investigations) | 1 | 0
Hepatic enzyme increased (Investigations) | 1 | 0
International normalised ratio increased (Investigations) | 1 | 0
Myocardial necrosis marker increased (Investigations) | 0 | 1
Oxygen saturation decreased (Investigations) | 0 | 1
Protein urine present (Investigations) | 0 | 1
Scan myocardial perfusion abnormal (Investigations) | 0 | 1
Troponin increased (Investigations) | 0 | 1
Urine albumin/creatinine ratio increased (Investigations) | 0 | 1
Vitamin B1 decreased (Investigations) | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 31 | 21
Hypoglycaemia (Metabolism and nutrition disorders) | 19 | 19
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 7 | 14
Hyperglycaemia (Metabolism and nutrition disorders) | 12 | 9
Dehydration (Metabolism and nutrition disorders) | 6 | 10
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 7 | 6
Hyperkalaemia (Metabolism and nutrition disorders) | 8 | 4
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 8 | 3
Obesity (Metabolism and nutrition disorders) | 5 | 6
Gout (Metabolism and nutrition disorders) | 3 | 6
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 6 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 3 | 1
Decreased appetite (Metabolism and nutrition disorders) | 2 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 2
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 1 | 1
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 2
Diabetic complication (Metabolism and nutrition disorders) | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1
Fluid overload (Metabolism and nutrition disorders) | 1 | 0
Hyperinsulinaemic hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 0
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0
Insulin-requiring type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Metabolic syndrome (Metabolism and nutrition disorders) | 0 | 1
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 37 | 38
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 7 | 17
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 8
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 7 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 5
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 7 | 4
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 2 | 5
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 3 | 4
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 5 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 4 | 2
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 2 | 3
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 | 1
Neuropathic arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 3
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 2 | 2
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 2
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 2
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 0 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0
Periarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 | 2
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 2
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 2
Vertebral foraminal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 1
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Back disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 0 | 1
Chondropathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Connective tissue inflammation (Musculoskeletal and connective tissue disorders) | 1 | 0
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Facet joint syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1
Fasciitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Femoroacetabular impingement (Musculoskeletal and connective tissue disorders) | 0 | 1
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 | 0
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint instability (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal ligament ossification (Musculoskeletal and connective tissue disorders) | 1 | 0
Spondylitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Tendon pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 26 | 30
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 7
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 7 | 7
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 7
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 5
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 5
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 5
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 6
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 6
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 3
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 2
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 6
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 4
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3
Laryngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 1
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 1
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 0
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Invasive lobular breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Hepatic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Intraductal papillary mucinous neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3
Prostate cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Benign breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Lip and/or oral cavity cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Metastases to peritoneum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Metastatic renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Metastatic squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Oesophageal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Papillary cystadenoma lymphomatosum (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Papillary renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Rectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Transitional cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Ureteral neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Adenocarcinoma of appendix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Adenoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Benign small intestinal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder cancer stage 0, with cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder transitional cell carcinoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bone cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Brain cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Chondrosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Chondrosarcoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Choroid melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colorectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colorectal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Dysplastic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Endometrial cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Epithelioid sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Essential thrombocythaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Follicular thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gallbladder adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gallbladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hodgkin's disease mixed cellularity stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hypergammaglobulinaemia benign monoclonal (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hypopharyngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Intestinal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Intraductal papillary-mucinous carcinoma of pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Laryngeal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lip neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung adenocarcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant ascites (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant mediastinal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant melanoma stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant palate neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant peritoneal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Melanoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to kidney (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to pleura (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Monoclonal gammopathy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Myelofibrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Myeloproliferative neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Neuroendocrine tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neuroendocrine tumour of the lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Oropharyngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Paranasal sinus neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Parathyroid tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Phaeochromocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pituitary tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pleomorphic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pleural neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prolactin-producing pituitary tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rectal cancer stage I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rectal cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal cell carcinoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal oncocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Salivary gland cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Small cell lung cancer extensive stage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Small intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Soft tissue sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma of the parotid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Synovial sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Testicular leiomyosarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Transitional cell carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 52 | 53
Cerebrovascular accident (Nervous system disorders) | 26 | 25
Syncope (Nervous system disorders) | 27 | 21
Transient ischaemic attack (Nervous system disorders) | 20 | 21
Carotid artery stenosis (Nervous system disorders) | 12 | 11
Cerebral infarction (Nervous system disorders) | 6 | 6
Diabetic neuropathy (Nervous system disorders) | 4 | 6
Seizure (Nervous system disorders) | 3 | 7
Cerebrovascular disorder (Nervous system disorders) | 4 | 3
Encephalopathy (Nervous system disorders) | 4 | 3
Headache (Nervous system disorders) | 3 | 4
Dizziness (Nervous system disorders) | 6 | 0
Hemiparesis (Nervous system disorders) | 2 | 4
Lacunar stroke (Nervous system disorders) | 1 | 5
Embolic stroke (Nervous system disorders) | 1 | 4
Lacunar infarction (Nervous system disorders) | 1 | 4
Presyncope (Nervous system disorders) | 2 | 3
Carotid artery occlusion (Nervous system disorders) | 4 | 0
Cerebral haemorrhage (Nervous system disorders) | 2 | 2
Lumbar radiculopathy (Nervous system disorders) | 3 | 1
Subarachnoid haemorrhage (Nervous system disorders) | 2 | 2
Altered state of consciousness (Nervous system disorders) | 3 | 0
Bell's palsy (Nervous system disorders) | 0 | 3
Cerebellar infarction (Nervous system disorders) | 2 | 1
Cerebellar stroke (Nervous system disorders) | 1 | 2
Cervical radiculopathy (Nervous system disorders) | 2 | 1
Haemorrhagic stroke (Nervous system disorders) | 2 | 1
Intracranial aneurysm (Nervous system disorders) | 2 | 1
Loss of consciousness (Nervous system disorders) | 3 | 0
Metabolic encephalopathy (Nervous system disorders) | 1 | 2
Sciatica (Nervous system disorders) | 0 | 3
Balance disorder (Nervous system disorders) | 1 | 1
Brain stem stroke (Nervous system disorders) | 1 | 1
Carotid arteriosclerosis (Nervous system disorders) | 0 | 2
Carpal tunnel syndrome (Nervous system disorders) | 2 | 0
Cognitive disorder (Nervous system disorders) | 2 | 0
Epilepsy (Nervous system disorders) | 1 | 1
Hypertensive encephalopathy (Nervous system disorders) | 0 | 2
Myelopathy (Nervous system disorders) | 2 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 1
Quadriplegia (Nervous system disorders) | 1 | 1
Radiculopathy (Nervous system disorders) | 1 | 1
Thrombotic stroke (Nervous system disorders) | 0 | 2
Toxic encephalopathy (Nervous system disorders) | 2 | 0
Amyotrophic lateral sclerosis (Nervous system disorders) | 0 | 1
Anosmia (Nervous system disorders) | 0 | 1
Aphasia (Nervous system disorders) | 1 | 0
Ataxia (Nervous system disorders) | 1 | 0
Basal ganglia haemorrhage (Nervous system disorders) | 0 | 1
Brain stem infarction (Nervous system disorders) | 0 | 1
Carotid artery aneurysm (Nervous system disorders) | 0 | 1
Carotid artery disease (Nervous system disorders) | 1 | 0
Carotid artery insufficiency (Nervous system disorders) | 1 | 0
Carotid sinus syndrome (Nervous system disorders) | 1 | 0
Cauda equina syndrome (Nervous system disorders) | 0 | 1
Central nervous system lesion (Nervous system disorders) | 0 | 1
Cerebellar syndrome (Nervous system disorders) | 1 | 0
Cerebral arteriosclerosis (Nervous system disorders) | 0 | 1
Cerebral ischaemia (Nervous system disorders) | 1 | 0
Cerebral microangiopathy (Nervous system disorders) | 1 | 0
Cerebrospinal fluid leakage (Nervous system disorders) | 0 | 1
Cerebrovascular insufficiency (Nervous system disorders) | 1 | 0
Cervical cord compression (Nervous system disorders) | 1 | 0
Chronic inflammatory demyelinating polyradiculoneuropathy (Nervous system disorders) | 1 | 0
Colloid brain cyst (Nervous system disorders) | 0 | 1
Coma (Nervous system disorders) | 0 | 1
Coordination abnormal (Nervous system disorders) | 0 | 1
Depressed level of consciousness (Nervous system disorders) | 1 | 0
Dysarthria (Nervous system disorders) | 1 | 0
Encephalomalacia (Nervous system disorders) | 0 | 1
Facial paralysis (Nervous system disorders) | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 1 | 0
Haemorrhagic transformation stroke (Nervous system disorders) | 1 | 0
Hemiplegia (Nervous system disorders) | 0 | 1
Hepatic encephalopathy (Nervous system disorders) | 1 | 0
Hydrocephalus (Nervous system disorders) | 0 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 0
Hypoglycaemic encephalopathy (Nervous system disorders) | 1 | 0
Hypoglycaemic seizure (Nervous system disorders) | 1 | 0
Hypotonia (Nervous system disorders) | 1 | 0
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 1 | 0
Intensive care unit acquired weakness (Nervous system disorders) | 0 | 1
Intracranial pressure increased (Nervous system disorders) | 0 | 1
Ischaemic cerebral infarction (Nervous system disorders) | 1 | 0
Lumbosacral radiculopathy (Nervous system disorders) | 0 | 1
Monoparesis (Nervous system disorders) | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 1
Nystagmus (Nervous system disorders) | 1 | 0
Ophthalmic migraine (Nervous system disorders) | 0 | 1
Optic neuritis (Nervous system disorders) | 0 | 1
Paraparesis (Nervous system disorders) | 1 | 0
Parkinson's disease (Nervous system disorders) | 1 | 0
Partial seizures (Nervous system disorders) | 1 | 0
Postresuscitation encephalopathy (Nervous system disorders) | 0 | 1
Psychomotor hyperactivity (Nervous system disorders) | 0 | 1
Restless legs syndrome (Nervous system disorders) | 0 | 1
Reversible cerebral vasoconstriction syndrome (Nervous system disorders) | 1 | 0
Spinal cord compression (Nervous system disorders) | 1 | 0
Spinal cord haematoma (Nervous system disorders) | 0 | 1
Spinal cord herniation (Nervous system disorders) | 0 | 1
Spinal cord infarction (Nervous system disorders) | 0 | 1
Status migrainosus (Nervous system disorders) | 0 | 1
Tension headache (Nervous system disorders) | 0 | 1
Transient global amnesia (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 1 | 0
Uraemic encephalopathy (Nervous system disorders) | 0 | 1
Vascular dementia (Nervous system disorders) | 0 | 1
Vascular parkinsonism (Nervous system disorders) | 0 | 1
Vertebral artery occlusion (Nervous system disorders) | 1 | 0
Vertebrobasilar insufficiency (Nervous system disorders) | 1 | 0
Vertebrobasilar stroke (Nervous system disorders) | 1 | 0
VIth nerve paralysis (Nervous system disorders) | 1 | 0
VIth nerve paresis (Nervous system disorders) | 1 | 0
Device malfunction (Product Issues) | 1 | 1
Device power source issue (Product Issues) | 1 | 1
Lead dislodgement (Product Issues) | 1 | 1
Device breakage (Product Issues) | 0 | 1
Device dislocation (Product Issues) | 1 | 0
Device electrical impedance issue (Product Issues) | 1 | 0
Device fastener issue (Product Issues) | 1 | 0
Device occlusion (Product Issues) | 0 | 1
Depression (Psychiatric disorders) | 3 | 4
Delirium (Psychiatric disorders) | 3 | 2
Anxiety (Psychiatric disorders) | 2 | 2
Major depression (Psychiatric disorders) | 2 | 2
Suicidal ideation (Psychiatric disorders) | 2 | 2
Disorientation (Psychiatric disorders) | 1 | 2
Mental status changes (Psychiatric disorders) | 2 | 1
Suicide attempt (Psychiatric disorders) | 1 | 2
Bipolar disorder (Psychiatric disorders) | 1 | 1
Confusional state (Psychiatric disorders) | 0 | 2
Schizophrenia (Psychiatric disorders) | 1 | 1
Conversion disorder (Psychiatric disorders) | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 0
Mental disorder (Psychiatric disorders) | 1 | 0
Panic attack (Psychiatric disorders) | 0 | 1
Post-traumatic stress disorder (Psychiatric disorders) | 0 | 1
Psychotic disorder (Psychiatric disorders) | 0 | 1
Sleep disorder (Psychiatric disorders) | 0 | 1
Substance-induced psychotic disorder (Psychiatric disorders) | 0 | 1
Suspected suicide (Psychiatric disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 66 | 42
Nephrolithiasis (Renal and urinary disorders) | 13 | 16
Chronic kidney disease (Renal and urinary disorders) | 11 | 6
Renal failure (Renal and urinary disorders) | 8 | 8
Urinary retention (Renal and urinary disorders) | 6 | 7
Ureterolithiasis (Renal and urinary disorders) | 4 | 7
Diabetic nephropathy (Renal and urinary disorders) | 9 | 1
Calculus urinary (Renal and urinary disorders) | 6 | 1
Haematuria (Renal and urinary disorders) | 5 | 2
Renal impairment (Renal and urinary disorders) | 3 | 4
Hydronephrosis (Renal and urinary disorders) | 3 | 2
End stage renal disease (Renal and urinary disorders) | 3 | 1
Proteinuria (Renal and urinary disorders) | 3 | 1
Urethral stenosis (Renal and urinary disorders) | 2 | 2
Calculus bladder (Renal and urinary disorders) | 1 | 2
Renal artery stenosis (Renal and urinary disorders) | 3 | 0
Renal cyst (Renal and urinary disorders) | 2 | 1
Urinary tract obstruction (Renal and urinary disorders) | 2 | 1
Bladder tamponade (Renal and urinary disorders) | 1 | 1
Nephrotic syndrome (Renal and urinary disorders) | 2 | 0
Renal colic (Renal and urinary disorders) | 2 | 0
Ureteric stenosis (Renal and urinary disorders) | 0 | 2
Azotaemia (Renal and urinary disorders) | 1 | 0
Bladder prolapse (Renal and urinary disorders) | 1 | 0
Cystitis haemorrhagic (Renal and urinary disorders) | 1 | 0
Dysuria (Renal and urinary disorders) | 0 | 1
Glomerulonephritis (Renal and urinary disorders) | 1 | 0
Haemorrhage urinary tract (Renal and urinary disorders) | 1 | 0
Hypertonic bladder (Renal and urinary disorders) | 0 | 1
Nephropathy toxic (Renal and urinary disorders) | 1 | 0
Nephrosclerosis (Renal and urinary disorders) | 1 | 0
Renal haematoma (Renal and urinary disorders) | 1 | 0
Renal mass (Renal and urinary disorders) | 0 | 1
Renal tubular injury (Renal and urinary disorders) | 1 | 0
Stag horn calculus (Renal and urinary disorders) | 0 | 1
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 | 0
Ureteric obstruction (Renal and urinary disorders) | 0 | 1
Urethral meatus stenosis (Renal and urinary disorders) | 1 | 0
Urinary bladder varices (Renal and urinary disorders) | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 17 | 13
Prostatitis (Reproductive system and breast disorders) | 0 | 4
Uterine polyp (Reproductive system and breast disorders) | 1 | 1
Acquired hydrocele (Reproductive system and breast disorders) | 1 | 0
Adnexa uteri mass (Reproductive system and breast disorders) | 0 | 1
Balanoposthitis (Reproductive system and breast disorders) | 0 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 1
Female genital tract fistula (Reproductive system and breast disorders) | 0 | 1
Penile haematoma (Reproductive system and breast disorders) | 0 | 1
Penile necrosis (Reproductive system and breast disorders) | 0 | 1
Uterine haemorrhage (Reproductive system and breast disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 23 | 15
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 22 | 16
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 27 | 9
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 15 | 14
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 | 10
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 5 | 9
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 | 8
Asthma (Respiratory, thoracic and mediastinal disorders) | 5 | 5
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 9
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 7 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 5
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pickwickian syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary cavitation (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Aorto-bronchial fistula (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoventilation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Nasal cavity mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Paraneoplastic pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pharyngeal cyst (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary sarcoidosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Vocal cord cyst (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Vocal cord polyp (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Vocal cord thickening (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Diabetic foot (Skin and subcutaneous tissue disorders) | 15 | 10
Skin ulcer (Skin and subcutaneous tissue disorders) | 9 | 10
Angioedema (Skin and subcutaneous tissue disorders) | 3 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 1
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 1
Cutaneous vasculitis (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Henoch-Schonlein purpura (Skin and subcutaneous tissue disorders) | 0 | 1
Necrotic angiodermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Prurigo (Skin and subcutaneous tissue disorders) | 0 | 1
Purpura (Skin and subcutaneous tissue disorders) | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1
Skin necrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Death of relative (Social circumstances) | 0 | 1
Housebound (Social circumstances) | 1 | 0
Cardiac pacemaker replacement (Surgical and medical procedures) | 1 | 0
Hysterosalpingo-oophorectomy (Surgical and medical procedures) | 1 | 0
Limb amputation (Surgical and medical procedures) | 0 | 1
Peripheral arterial occlusive disease (Vascular disorders) | 37 | 60
Hypertensive crisis (Vascular disorders) | 13 | 17
Hypertension (Vascular disorders) | 19 | 10
Aortic stenosis (Vascular disorders) | 12 | 9
Deep vein thrombosis (Vascular disorders) | 12 | 6
Hypotension (Vascular disorders) | 8 | 10
Peripheral ischaemia (Vascular disorders) | 5 | 8
Peripheral artery stenosis (Vascular disorders) | 5 | 6
Orthostatic hypotension (Vascular disorders) | 5 | 5
Peripheral artery occlusion (Vascular disorders) | 5 | 5
Peripheral artery thrombosis (Vascular disorders) | 3 | 7
Aortic aneurysm (Vascular disorders) | 5 | 4
Hypertensive emergency (Vascular disorders) | 5 | 4
Iliac artery stenosis (Vascular disorders) | 5 | 4
Extremity necrosis (Vascular disorders) | 3 | 5
Intermittent claudication (Vascular disorders) | 6 | 2
Peripheral artery aneurysm (Vascular disorders) | 3 | 3
Peripheral vascular disorder (Vascular disorders) | 3 | 3
Haematoma (Vascular disorders) | 2 | 3
Circulatory collapse (Vascular disorders) | 2 | 2
Hypertensive urgency (Vascular disorders) | 3 | 1
Arteriosclerosis (Vascular disorders) | 2 | 1
Diabetic vascular disorder (Vascular disorders) | 1 | 2
Dry gangrene (Vascular disorders) | 1 | 2
Hypovolaemic shock (Vascular disorders) | 1 | 2
Venous thrombosis (Vascular disorders) | 2 | 1
Arterial thrombosis (Vascular disorders) | 0 | 2
Distributive shock (Vascular disorders) | 1 | 1
Embolism arterial (Vascular disorders) | 2 | 0
Pelvic venous thrombosis (Vascular disorders) | 2 | 0
Shock haemorrhagic (Vascular disorders) | 1 | 1
Thrombosis (Vascular disorders) | 1 | 1
Varicose vein (Vascular disorders) | 0 | 2
Aneurysm (Vascular disorders) | 1 | 0
Aortic aneurysm rupture (Vascular disorders) | 0 | 1
Aortic arteriosclerosis (Vascular disorders) | 0 | 1
Aortic dissection (Vascular disorders) | 1 | 0
Aortic occlusion (Vascular disorders) | 0 | 1
Aortic thrombosis (Vascular disorders) | 0 | 1
Arterial insufficiency (Vascular disorders) | 0 | 1
Arterial occlusive disease (Vascular disorders) | 0 | 1
Arterial stenosis (Vascular disorders) | 0 | 1
Femoral artery aneurysm (Vascular disorders) | 1 | 0
Haemorrhagic infarction (Vascular disorders) | 1 | 0
Iliac artery dissection (Vascular disorders) | 1 | 0
Iliac artery occlusion (Vascular disorders) | 0 | 1
Infarction (Vascular disorders) | 1 | 0
Ischaemia (Vascular disorders) | 0 | 1
Ischaemic limb pain (Vascular disorders) | 1 | 0
Leriche syndrome (Vascular disorders) | 0 | 1
Neurogenic shock (Vascular disorders) | 0 | 1
Phlebitis (Vascular disorders) | 0 | 1
Subclavian artery stenosis (Vascular disorders) | 1 | 0
Thromboangiitis obliterans (Vascular disorders) | 1 | 0
Thrombophlebitis (Vascular disorders) | 1 | 0
Varicose ulceration (Vascular disorders) | 0 | 1
Vasculitis (Vascular disorders) | 1 | 0
Venous stenosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pemafibrate (N=5264) | Placebo (N=5274)
Diarrhoea (Gastrointestinal disorders) | 308 | 343
Urinary tract infection (Infections and infestations) | 417 | 461
COVID-19 (Infections and infestations) | 361 | 377
Nasopharyngitis (Infections and infestations) | 358 | 354
Coronavirus infection (Infections and infestations) | 221 | 265
Influenza (Infections and infestations) | 251 | 290
Diabetes mellitus (Metabolism and nutrition disorders) | 738 | 677
Arthralgia (Musculoskeletal and connective tissue disorders) | 417 | 454
Back pain (Musculoskeletal and connective tissue disorders) | 311 | 355
Headache (Nervous system disorders) | 227 | 265
Diabetic nephropathy (Renal and urinary disorders) | 358 | 343
Hypertension (Vascular disorders) | 683 | 664

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (4):
  • Study Protocol: Initial (2016-11-16): https://cdn.clinicaltrials.gov/large-docs/92/NCT03071692/Prot_000.pdf
  • Study Protocol: Amdt. 1 (2017-03-27): https://cdn.clinicaltrials.gov/large-docs/92/NCT03071692/Prot_001.pdf
  • Study Protocol: Amdt. 2 (2020-03-18): https://cdn.clinicaltrials.gov/large-docs/92/NCT03071692/Prot_002.pdf
  • Statistical Analysis Plan (2022-10-24): https://cdn.clinicaltrials.gov/large-docs/92/NCT03071692/SAP_003.pdf